

## **Statistical Analysis Plan**

SAP Text Version Number: Final Version

SAP Text Date: 19-Jan-2024

Sponsor Name: Galderma S.A./Galderma R&D, LLC

Protocol Number: RD.06.SPR.203890

Protocol Title: A Double-Blind, Placebo-Controlled, Randomized Study to Assess the Durability of Effect

and Safety of Nemolizumab for 24 Weeks in Subjects with Prurigo Nodularis

#### **Protocol Version and Date:**

V1.0, 20-Jul-2021

V2.0, 12-Dec-2022

V2.0, 22-Mar-2022 - For Germany

V3.0, 12-Dec-2022 - For Germany

**Authors: PPD** 

#### **Notice of Confidential and Proprietary Information:**

The information contained in this document is confidential belonging to Galderma S.A./Galderma R&D, LLC. Acceptance of this document constitutes agreement by the recipient that no information contained herein will be published or disclosed without prior written authorization from an official of Galderma S.A./Galderma R&D, LLC. However, this document may be disclosed to appropriate Institutional Review Board and Ethics Committees or duly authorized representatives of a national regulatory authority under the condition that they are requested to keep it confidential. In the event of an actual or suspected breach of this obligation, **CCI** should be notified promptly.

# **Revision History**

| Version # | Date<br>(DD-Mmm-YYYY) | Document Owner | Revision Summary |
|---|---|---|---|
| 1.0 | 11-Jan-2024 | PPD | Final ∀ersion |
| 2.0 | 19-Jan2024 | PPD | <ul> <li>Protocol version update on the title page</li> <li>Sample size section 4.3 updated with protocol Version 3.0</li> </ul> |

I confirm that I have reviewed this document and agree with the content.

| Approvals | | |
|---|---|---|
| CCI | | |
| PPD | PPD | |
| Name, Title<br>Lead Biostatistician | Signature | Date (DD-Mmm-<br>YYYY) |
| PPD | PPD | |
| Name, Title Senior Reviewing Biostatistician | Signature | Date (DD-Mmm-<br>YYYY) |
| Galderma S.A./Ga | alderma R&D, LLC Approval | |
| PPD | PPD | |
| Name, Title<br>Sponsor Contact | Signature | Date (DD-Mmm-<br>YYYY) |

## **Table of Contents**

| Revi | sion His | story | 2 |
|------|----------|---------------------------------------|----|
| Арр | rovals | | 3 |
| 1. | Glossa | ary of Abbreviations | 7 |
| 2. | Purpo | se | 12 |
| | 2.1. | Responsibilities | 12 |
| | 2.2. | Timings of Analyses | 12 |
| 3. | Study | Objectives | 13 |
| | 3.1. | Primary Objective | 13 |
| | 3.2. | Secondary Objectives | 13 |
| 4. | Study | Details/Design | 14 |
| | 4.1. | Brief Description | 14 |
| | 4.2. | Subject Selection | 18 |
| | | 4.2.1. Inclusion Criteria | 18 |
| | | 4.2.2. Exclusion Criteria | 18 |
| | 4.3. | Determination of Sample Size | 18 |
| | 4.4. | Treatment Assignment and Blinding | 18 |
| | 4.5. | Administration of Study Medication | 20 |
| | 4.6. | Study Procedures and Flowchart | 21 |
| 5. | Endpo | oints | 25 |
| | 5.1. | Primary Efficacy Endpoints | 25 |
| | 5.2. | Secondary Efficacy Endpoints | 25 |
| | 5.3. | Safety Endpoints | 25 |
| 6. | Analys | sis Sets | 27 |
| | 6.1. | Intent-to-Treat Population | 27 |
| | 6.2. | Safety Population | 27 |
| | 6.3. | Proof of Exposure Analysis Population | 27 |
| | 6.4. | Per-Protocol Population | 27 |
| | 6.5. | Protocol Deviations | 27 |
| 7. | Estima | ands | 29 |
| 8. | Gener | al Aspects for Statistical Analysis | 31 |
| | 8.1. | General Methods | 31 |

| | 8.2. | Key De | finitions | 31 |
|---|---|---|---|---|
| | 8.3. | Missing | Data | 32 |
| | 8.4. | Visit Wi | ndows | 33 |
| | 8.5. | Subgrou | ups | 35 |
| 9. | Demo | graphic, ( | Other Baseline Characteristics and Medication | 36 |
| | 9.1. | Subject | Disposition and Withdrawals | 36 |
| | 9.2. | Demog | raphic and Baseline Disease Characteristics | 36 |
| | 9.3. | Medical | History | 37 |
| | 9.4. | Medical | and Surgical Procedure | 37 |
| | 9.5. | Medicat | tion | 38 |
| | 9.6. | Extent of | of Exposure | 39 |
| | 9.7. | Treatme | ent Compliance | 39 |
| 10. | Efficad | cy | | 40 |
| | 10.1. | Primary | Efficacy Endpoints | 40 |
| | | 10.1.1. | Primary Analysis of Primary Efficacy Endpoint | 40 |
| | | 10.1.2. | Sensitivity Analyses of Primary Efficacy Endpoint | 41 |
| | 10.2. | Second | ary Efficacy Endpoints | 41 |
| | | 10.2.1. | Investigator's Global Assessment (IGA) | 43 |
| | | 10.2.2. | Pruritus Numeric Rating Scale (NRS) | 43 |
| | | 10.2.3. | Sleep Disturbance Numeric Rating Scale (SD NRS) | 45 |
| | | 10.2.4. | Dermatology Life Quality Index | 46 |
| 11. | Pharm | nacokinet | ics | 47 |
| | 11.1. | Pharma | cokinetic Concentration Presentation | 47 |
| 12. | Immur | nogenicity | y | 48 |
| 13. | Safety | <i>'</i> | | 49 |
| | 13.1. | Adverse | e Events | 49 |
| | 13.2. | Laborat | ory Evaluations | 52 |
| | | 13.2.1. | Clinical Laboratory Evaluations | 52 |
| | | 13.2.2. | Pregnancy Testing | 53 |
| | | 13.2.3. | Virology and TB Testing | 54 |
| | 13.3. | Vital Sig | gns | 54 |
| | 13.4 | ECG | | 55 |

| | 13.5. | Physical | Examination | 55 |
|-----|---------|-------------|-----------------------------------|----|
| | 13.6. | Respirat | ory Assessments | 56 |
| | | 13.6.1. | Asthma Control Test | 56 |
| | | 13.6.2. | Respiratory Examination | 56 |
| | | 13.6.3. | Peak Expiratory Flow | 57 |
| 14. | Chang | es from A | Analysis Planned in Protocol | 58 |
| 15. | Progra | mming C | onsiderations | 59 |
| | 15.1. | General | Considerations | 59 |
| | 15.2. | Table, F | igure, and Listing Format | 59 |
| | | 15.2.1. | General | 59 |
| | | 15.2.2. | Headers | 60 |
| | | 15.2.3. | Display Titles | 60 |
| | | 15.2.4. | Column Headers | 60 |
| | | 15.2.5. | Body of the Data Display | 61 |
| | | 15.2.6. | Footnotes | 63 |
| 16. | Quality | / Control | | 65 |
| 17. | Index | of Tables | | 66 |
| 18. | Index | of Figures | 5 | 81 |
| 19. | Index | of Listings | S | 82 |
| 20. | Appen | dices | | 85 |
| | 20.1. | Example | SAS Code | 85 |
| | 20.2. | Potentia | lly Clinically Significant Ranges | 87 |

#### 1. **Glossary of Abbreviations**

| Abbreviation | Description |
|--------------|-----------------------------------|
| ACT | Asthma Control Test |
| ADA | Anti-Drug Antibodies |
| ADaM | Analysis Dataset Model |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ALP | Alkaline Phosphatase |
| ALT | Alanine Aminotransferase |
| ANCOVA | Analysis of Covariance |
| AP | Average Pruritus |
| AST | Aspartate Aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BDRM | Blind Data Review Meeting |
| BMI | Body Mass Index |
| СНМР | Committee for Medicinal Products |
| CI | Confidence Interval |
| СМН | Cochran-Mantel-Haenszel |
| COVID-19 | Coronavirus Disease-19 |
| CRA | Clinical Research Associate |
| CRF | Case Report Form |
| CRO | Contract Research Organization |
| CS | Clinical Significant |
| CSR | Clinical Study Report |
| CTMS | Clinical Trial Management System |
| CV | Coefficient of Variation |

| Abbreviation | Description |
|--------------|-------------------------------------------|
| D | Depression |
| DBL | Data Base Lock |
| DCS | Dual-Chamber Syringe |
| DD | Drug Dictionary |
| DLQI | Dermatology Life Quality Index |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| ET | Early Termination |
| FSH | Follicle-Stimulating Hormone |
| HADS | Hospital Anxiety and Depression Scale |
| HBcAb | Hepatitis B core Antibody |
| HBsAg | Hepatitis B surface Antigen |
| HCV | Hepatitis C Virus |
| HDL | High-Density Lipoproteins |
| HIV | Human Immunodeficiency Virus |
| IAC | Independent Adjudication Committee |
| IB | Investigator's Brochure |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IGA | Investigator Global Assessment |
| IL-31 | Interleukin-31 |
| IRT | Interactive Response Technology |
| ITT | Intent-to-Treat |
| IVRS | Interactive Voice Response System |

| Abbreviation | Description |
|--------------|----------------------------------------------|
| IWRS | Interactive Web Response System |
| LDL | Low-Density Lipoproteins |
| LLN | Lower Limit of Normal |
| LTE | Long-Term Extension |
| LSMeans | Least Squares Means |
| MAR | Missing at Random |
| MCMC | Markov chain Monte Carlo |
| MedDRA | Medical Dictionary for Regulatory Activities |
| МІ | Multiple Imputation |
| min | Minutes |
| MMRM | Mixed-Effect Models for Repeated Measures |
| MSD | Morning Sleep Diary |
| N/A | Not Applicable |
| NAb | Neutralizing Antibodies |
| NCS | Not Clinical Significant |
| NK | Neurokinin |
| NRS | Numeric Rating Scale |
| ОС | Observed Case |
| PCR | Polymerase Chain Reaction |
| PD | Pharmacodynamics |
| PDF | Portable Document Format |
| PEF | Peak Expiratory Flow |
| PK | Pharmacokinetic |
| PN | Prurigo Nodularis |
| POE | Proof of Exposure |

| Abbreviation | Description |
|--------------|-------------------------------------------|
| PP NRS | Peak Pruritus Numeric Rating Scale |
| PP | Peak Pruritus |
| PPS | Per-Protocol Set |
| PT | Preferred Term |
| Q1 | 1st Quartile |
| Q3 | 3d Quartile |
| Q4W | Every 4 Weeks |
| QC | Quality Control |
| QoL | Quality of Life |
| RNA | Ribonucleic Acid |
| RTSM | Randomization and Trial Supply Management |
| SAE | Serious Adverse Event |
| SAF | Safety Population |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis System |
| sc | Subcutaneous |
| SD | Standard Deviation |
| SD NRS | Sleep Disturbance Numeric Rating Scale |
| SDTM | Study Data Tabulation Model |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| ТВ | Tuberculosis |
| TEAE | Treatment-Emergent Adverse Event |
| TFL | Table, Figure and Listing |
| TMF | Trial Master File |

Statistical Analysis Plan for Interventional Studies
Sponsor: Galderma S.A./Galderma R&D, LLC; Protocol No.: RD.06.SPR.203890

| Abbreviation | Description |
|--------------|---------------------------|
| ULN | Upper Limit of Normal |
| UPT | Urine Pregnancy Test |
| US | United States |
| W | Week |
| WHO | World Health Organization |

2. Purpose

The purpose of this statistical analysis plan (SAP) is to ensure that the data listings, summary tables and

figures which will be produced, and the statistical methodologies that will be used, are complete and

appropriate to allow valid conclusions regarding the study objectives. The planned analyses identified in

this SAP will be included in regulatory submissions and/or future manuscripts. Exploratory analyses not

identified or defined in this SAP may be performed to support the clinical development program. Any post-

hoc or unplanned analyses performed and not identified in this SAP will be documented in the respective

clinical study report (CSR).

2.1. Responsibilities

will perform the statistical analyses and is responsible for the production and quality control

of all tables, figures and listings.

2.2. Timings of Analyses

The final analysis may be carried out once all subjects have completed the final study visit or terminate

early from the study. No personnel directly involved with the conduct of the study shall have access to the

unblinded data before the completion of the trial in order to avoid introducing bias to the remaining study

data.

An interim analysis may be conducted for the submission of the regulatory registration of nemolizumab.

An independent data monitoring committee (IDMC) will review and monitor subject safety throughout the

study, and an independent adjudication committee (IAC) will review all asthma-related adverse events

throughout the study. Details on the IDMC and IAC, including the plan of analysis for outputs; the

composition of the committees; and the procedures, roles, responsibilities, and communications are

provided in the respective IDMC (v1.0, dated 24-Aug-2020) and Appendix 2 of IAC charters (v1.0, dated

27-Aug-2020).

## 3. Study Objectives

### 3.1. Primary Objective

To assess the long-term durability of response over a 24-week period following withdrawal of nemolizumab in subjects with Pruigo Nodularis(PN) who previously responded to treatment in the Long-Term Extension (LTE) study RD.06.SPR.202699.

## 3.2. Secondary Objectives

To assess the safety of nemolizumab compared to placebo over a 24-week period in subjects with PN who previously responded to treatment in the LTE study.

4. Study Details/Design

4.1. Brief Description

This is a Phase 3b multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the durability of response and safety of nemolizumab in adult subjects who participated in the nemolizumab PN LTE study (RD.06.SPR.202699) and achieved a clinical response (i.e., IGA score of 0 or 1 and ≥4-point improvement in weekly average of PP NRS score from baseline of the lead-in study) at

Week 52 of the LTE study.

Subjects who agree to enroll in this study must do so at the time of completion of the Week 52 visit in the LTE study (RD.06.SPR.202699) to prevent any lapse in study treatment. After the Week 52 visit of the LTE study is complete, approximately 100 subjects who choose to enter this study will be randomized 1:1 to receive either 1 or 2 injections of nemolizumab or placebo, stratified by dosing regimen. Subjects will continue to receive the same dosing regimen received in the LTE study (i.e., 1 or 2 SC injections of study

drug administered every 4 weeks [Q4W]). Subjects with a body weight <90 kg in LTE study will receive a

30-mg dose. Subjects weighing ≥90 kg in the LTE study will receive a 60-mg dose.

Subjects' participation in the study will be up to approximately 32 weeks. The study consists of a 24-week

treatment period and an 8-week follow-up period (12 weeks after their last study drug injection at Week 20).

Relapse is defined as an increase in (weekly average of the) PP NRS score ≥4 points from baseline or an increase in IGA score ≥ 2 from baseline at any point during the study. If a subject meets the criteria for relapse, then the subject may be considered for re-entry into the LTE study (RD.06.SPR.202699). Refer to

Figure 4-1 for subject transition between studies 202699 and 203890.

Figure 4-1: Subject Transition between Studies 202699 and 203890



\*Clinical responder is defined as a subject with an Investigator Global Assessment (IGA) score= 0 or 1 and improvement in Peak Pruritus Numeric Rating Scale (PP NRS) score of ≥4 points from baseline of the leadin study at Week 52 visit of the LTE study. Note: Lead-in study baseline is defined as baseline PP NRS score in the Phase 3 studies RD.06.SPR.202685 or RD.06.SPR.203065 for subjects who rolled over into the LTE from these studies. For subjects who entered the LTE study from the Phase 2 study RD.03.SPR.115828, the baseline PP NRS score at entry into the LTE study RD.06.SPR.202699 will be used.

\*\* Relapse is defined as an increase in weekly average of PP NRS score ≥4 points from baseline or an increase in IGA score ≥2 from baseline at any point during the study. Subjects who relapse at any point during the treatment period or who complete through Week 24 are eligible for LTE re-entry.

#### **Baseline Assessment**

After signing the informed consent form (ICF), all subjects will be evaluated for study participation, based on eligibility criteria. The study assessments at the time of completion of the Week 52 visit from the PN LTE lead-in study RD.06.SPR.202699 will be used as baseline assessments for the current study.

#### **Treatment Period**

Eligible subjects will be randomized to receive either 1 or 2 injections of nemolizumab or placebo according to their dosage group in the LTE study, as assigned by interactive response technology (IRT). Study drug

This document is confidential.

Filing requirements: TMF

will then be administered Q4W for 24 weeks with final dose administered at Week 20.

Refer to the below table for summary of the study treatment.

| LTE Lead-in Study | Lead-in Study Assigned | Dose Q4W for 24 weeks <sup>a</sup> |
|---|---|---|
| | Treatment | |
| | Nemolizumab | Blinded |
| | 30 mg | Nemolizumab 30 mg |
| | (1 injection) | (1 injection) |
| | | Blinded Placebo |
| | | (1 injection) |
| RD.06.SPR.202699 | | |
| 112.00.0111.202000 | Nemolizumab | Blinded |
| | 2 x 30 mg | Nemolizumab 2 x 30 mg |
| | (2 injections) | (2 injections) |
| | | Blinded 2 x Placebo |
| | | (2 injections) |

Abbreviation: LTE = long-term extension; Q4W = every 4 weeks.

Clinical assessments will occur according to the Schedule of Assessments in the protocol through the Week 24 visit.

If a subject meets the criteria for relapse at any point, the subject will exit the study and re-enter the LTE study (see Figure 4-1). Subjects who exit the study before Week 24 should complete an early termination (ET) visit. Subjects who complete the study through Week 24 are eligible to re-enroll in the LTE study.

Subjects who prematurely discontinue study drug for reasons other than relapse will be encouraged to complete the scheduled study visits. These subjects will only be eligible for re-enrollment in the LTE study if they continue with study visits through Week 24.

Subjects who discontinue the study for reasons other than relapse before Week 24 or who will not continue nemolizumab treatment in the LTE study should complete a follow-up visit, 12 weeks (±7 days) after the last study drug injection.

#### Follow-up Period

<sup>&</sup>lt;sup>a</sup> Dose will be assigned based on dose received in LTE lead-in study

A follow-up visit will be conducted 8 weeks (±7 days) after completing the treatment period and/or 12 weeks (±7 days) after the last study drug injection for all subjects who will not continue nemolizumab treatment in the LTE study. Twelve weeks corresponds to approximately 5 half-lives of nemolizumab when administered subcutaneously Q4W at the doses used in this study.

An overview of the study is presented in Figure 4-2.

Figure 4-2: Study Design



\*Clinical responder is defined as a subject with an Investigator Global Assessment (IGA) score= 0 or 1 and improvement in Peak Pruritus Numeric Rating Scale (PP NRS) score of ≥4 points from baseline of the leadin study at Week 52 visit of the LTE study. Note: Lead-in study baseline is defined as baseline PP NRS score in the Phase 3 studies RD.06.SPR.202685 or RD.06.SPR.203065 for subjects who rolled over into the LTE from these studies. For subjects who entered the LTE study from the Phase 2 study RD.03.SPR.115828, the baseline PP NRS score at entry into the LTE study RD.06.SPR.202699 will be used.

\*\* Relapse is defined as an increase in weekly average of PP NRS score ≥4 points from baseline or an


increase in IGA score ≥2 from baseline at any point during the study. Subjects who relapse at any point

during the treatment period or who complete through Week 24 are eligible for LTE re-entry.

Abbreviations: BL = baseline; LTE = long-term extension; R = randomization; W = week.

The end of the study will be the last subject's last visit as indicated in the Schedule of Assessments (Table

4-1).

4.2. Subject Selection

Eligible subjects for this clinical study will be adults who participated in the prior nemolizumab PN LTE study

(RD.06.SPR.202699) with uninterrupted dosing for 3 months before the Week 52 visit and achieved a

clinical response (i.e., IGA score of 0 or 1 and ≥4-point improvement in weekly average of PP NRS score

from baseline of the lead-in study) at Week 52. By randomizing subjects from the PN LTE study who

achieved a current clinical response to nemolizumab to either nemolizumab or placebo treatment arms, the

durability of the response to nemolizumab following discontinuation of active treatment (i.e., in the placebo

treatment arm) can be measured. This will be done to understand how long the effects of nemolizumab

treatment are expected to last in controlling signs and symptoms of PN when treatment is removed.

Subjects who experienced an AE during their participation in the prior lead-in study that in the opinion of

the Investigator could indicate that continued treatment with nemolizumab might present an unreasonable

risk for the subject are ineligible. Furthermore, subjects must not use restricted topical and systemic

treatments, including rescue therapy, within 6 months of the Week 52 visit in the PN LTE study.

4.2.1. Inclusion Criteria

For a detailed description of subject's inclusion criteria see protocol Section 8.1.

4.2.2. Exclusion Criteria

For a detailed description of subject's exclusion criteria see protocol Section 8.2.

4.3. Determination of Sample Size

No formal sample size calculations were performed for this study. The sample size will be based on the

sample size and the actual response rate of the LTE study. Based on the current assumption, it is expected

that approximately 40 subjects will be randomized.

4.4. Treatment Assignment and Blinding

Upon confirmation of eligibility for a given subject to participate in the study, a unique randomization number

will be assigned to that subject via Interactive Response Technology (IRT).

Statistical Analysis Plan for Interventional Studies


The randomization number for a given subject will be used to identify the treatment arm the subject will be

assigned to.

Subjects will be randomized in a 1:1 ratio to receive treatment of either Nemolizumab (CD14152) or

placebo. The randomization scheme will be stratified by dosing regimen (1 or 2 injections) using the IRT

system.

All attempts will be made to keep the study center staff and subjects blinded throughout the study. Members

of the study center staff, including those responsible for dual-chamber syringe (DCS) preparation, will not

have access to the randomized treatment assignment.

To ensure double-blind administration of study drug, the study center pharmacist(s) or other qualified

personnel will prepare all Nemolizumab (CD14152) or placebo treatments, according to the current version

of the pharmacy manual and assigned DCS provided by the IRT system.

As there may be detectable differences between active and placebo during the reconstitution process, the

DCS is delivered for injection after the reconstitution is complete. The pharmacist (or other qualified

personnel) preparing study drug should not be involved with any study assessments and should not discuss

any aspects of study drug reconstitution with the subject or study staff involved in subject interviews or

study assessments.

To maintain the integrity of the study blinding, the bioanalytical laboratory staff who process/analyze the

anti-drug antibody (ADA) samples will not provide any information to the Sponsor, CRO, or investigational

study center personnel directly involved with the ongoing conduct of the study that may lead to unblinding

during the ongoing study. ADA results will be released by the bioanalytical laboratory after data base lock

(DBL).

Unblinding of a subject's individual treatment code should occur only in case of a medical emergency or in

the event of a serious medical condition that necessitates identification of the study drug for the welfare of

that subject, as judged by the investigator. The emergency unblinding process utilizes IRT to allow the

investigator to have unrestricted, immediate, and direct access to the subject's individual study treatment.

When possible (i.e., when the health of the subject is not immediately at risk), the investigator or sub-

investigator is encouraged to consult with the medical monitor and the Sponsor before breaking the blind.

If emergency unblinding is required:

Only the investigator will make the decision to unblind the treatment assignment.

Only the affected subject will be unblinded.

Statistical Analysis Plan for Interventional Studies


The IRT system will provide the treatment assignment to the investigator.

Refer to the Randomization and Trial Supply Management (RTSM) User Guide for information on the steps

for breaking the blind in the IRT system.

When the blinding code is broken, the reason must be fully documented. If the code is broken by the

investigator, the subject must be withdrawn from the study and must also be appropriately followed for a

minimum of 12 weeks after the last dose of study drug.

The reporting requirements for unblinding are the same for reporting an SAE. See also Section 12.7.4 of

protocol.

The randomization code will remain blinded to all study sites and study team members until completion of

the study and after the study database has been locked.

An independent unblinded team will perform unblinded analysis at the time of interim analysis. Further

details are provided in unblinding plan.

The IDMC will review data at periodic intervals throughout the study as defined in the IDMC charter. The

IDMC charter will specify the procedures for unblinding to ensure treatment assignment remains

undisclosed to all individuals involved in the direct execution and management of the study until the final

database is locked.

4.5. Administration of Study Medication

"Study drug" or "study medication" refers to nemolizumab or placebo drug product for purposes of this

double-blind study. The list of excipients is detailed in the Investigator's Brochure(IB).

Study drug will be provided as lyophilized powder for solution for injection for SC use only after

reconstitution in a pre-filled, single-use, dual-chamber syringe (DCS).

The DCS is a self-contained system that holds the lyophilized nemolizumab or placebo and solution (sterile

water) for reconstitution, separately. The concentration of nemolizumab in the DCS will be 61.5 mg/mL

once reconstituted (volume of 0.49 mL per injection).

Subjects will receive nemolizumab or placebo according to their dosage group (1 or 2 SC injections) in the

LTE study, as assigned by IRT Q4W.

Subjects will have the option to self-inject study drug while at the study center under staff supervision.

Subjects will be trained on injecting the study drug and will be allowed to inject study drug following

appropriate training. If the subject does not wish to perform the injections, study staff can administer study drug at each visit.

## 4.6. Study Procedures and Flowchart

See Table 4-1 for study procedures.

Table 4-1: Schedule of Assessments

| | Baseline <sup>a</sup> | Treatment Period | | | | | | FU | ET | Unscheduled |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | | |
| Week | W0 (Day 1) | W4 | W8 | W12 | W16 | W20 | W24 | W32 | if applicable <sup>b</sup> | if<br>applicable ° |
| Visit Window (days) | | ±1 | ±3 | ±3 | ±3 | ±5 | ±5 | ±7 | | |
| ICF <sup>a</sup> | X | | | | | | | | | |
| Inclusion/exclusion | X | | | | | | | | | |
| Demographics | X | | | | | | | | | |
| Medical history, previous | | | | | | | | | | |
| therapies and | X | | | | | | | | | |
| procedures, smoking | | | | | | | | | | |
| status Patient-Reported Outco | mes | <u> </u> | | | <u> </u> | ļ | <u> </u> | | | |
| PP NRS/ SD NRS d.e | X | | | | | | | | X | (X) |
| DLQI e | Χ | 1 | 1 | 1 | X | I | X | $\vdash$ | X | (X) |
| Efficacy Assessments | | | | | <u> </u> | <u> </u> | <u> </u> | | ļ., | V-7 |
| IGA | Х | X | X | X | Х | Х | Х | ı | x | (X) |
| Safety Assessments | Λ | <u> ^</u> | ļ^ | <u> ^</u> | <u> ^</u> | <u> ^</u> | <u> ^</u> | <u> </u> | <u> ^</u> | (74) |
| ACT e.f | Х | X | X | Х | Х | Х | Х | Х | X | (X) |
| Respiratory examination | X | Χg | Χg | X | Χg | Χg | X | X | X | (X) |
| PEF testing | X | Χg | Χg | X | Χg | Χg | X | X | X | (X) |
| Vital signs h | X | X | X | X | X | X | X | X | X | (X) |
| | | | ^ | + | ^ | ^ | _ | - | | |
| Full physical examination | X | | | X | | | X | X | X | (X) |
| Symptom-directed | | | | | | | | | | |
| physical examination | | X | X | | X | X | | | | |
| Height | X | - | | | | | | - | | (X) |
| Weight | X | ├ | | | - | - | X | - | X | (X) |
| 12-lead ECG i | X | ╁ | | 1 | _ | | X | _ | X | |
| Contraceptive | | <del> </del> | | | <del> </del> | - | ^ | <del> </del> | ^ | (X) |
| counseling | X | | | | | | | | | (X) |
| Adverse events e | X | Х | Х | Х | Х | X | Х | Х | Х | (X) |
| Concomitant therapies | | 1 | | | | <u> </u> | t | | | |
| and procedures e | Х | X | Х | х | Х | X | X | X | х | (X) |
| · | | <u> </u> | | | <u> </u> | | | <u> </u> | | |
| Laboratory Assessment | is | | | | | , | | | , | |
| Blood samples for | | | | | | | | l, | | 00 |
| hematology and clinical | X | | | X | | | X | X | | (X) |
| chemistry <sup>j</sup> | | ļ | | | <u> </u> | | | | ļ | |
| Urinalysis | Х | | | Х | | | X | X | | (X) |
| Urine pregnancy test <sup>k</sup> | Х | X | X | Х | X | Х | Х | X | x | (X) |

| | Baseline <sup>a</sup> | Treatment Period | | | | FU | ET | Unscheduled | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | | if |
| Week | W0 (Day 1) | W4 | W8 | W12 | W16 | W20 | W24 | W32 | if applicable <sup>b</sup> | applicable ° |
| Visit Window (days) | | ±1 | ±3 | ±3 | ±3 | ±5 | ±5 | ±7 | | |
| FSH1 | X | | | | | | | | | (X) |
| Blood sample for virology<br>(HIV, Hepatitis B and C | | | | | | | | | | (X) |
| Blood sample for TB test | | | | | | | | | | (X) |
| POE & Immunogenicity | | | • | • | , | • | • | • | | |
| Blood sample for POE °. | х | | | | | | x | | х | (X) |
| Blood sample for ADA c, m | Х | | | | | | x | | х | (X) |
| Study Drug Administration | | | | | | | | | | |
| Randomization | Х | | | | | | | | | |
| Study drug injection <sup>n, o, p,</sup> | Х | x | х | х | x | x | | | | (X) |

ACT = Asthma Control Test; ADA = anti-drug antibody; AE = adverse event; DLQI = Dermatology Life Quality Index; ECG = electrocardiogram; ET = early termination; FSH = follicle-stimulating hormone; FU = follow-up; HIV = human immunodeficiency virus; ICF = informed consent form; IGA = Investigator Global Assessment; LTE = long-term extension; PEF = peak expiratory flow; POE = proof of exposure; PP NRS= peak pruritus numeric rating scale; SD NRS= sleep disturbance numeric rating scale; TB = tuberculosis; UPT = urine pregnancy test; V = visit; W = week.

- a) After signing the ICF, all subjects will be evaluated for study participation, based on eligibility criteria. The Week 52 study assessments from the LTE lead-in study RD.06.SPR.202699 will be used as baseline assessments for the current study.
- b) Subjects who relapse or discontinue prematurely (before the Week 24 visit) should complete an ET visit. If the subject discontinues for reasons other than relapse before Week 24, or will not continue with nemolizumab treatment in the LTE study, a follow-up visit should also be completed, 12 weeks (±7 days) after the last study drug injection.
- c) Assessments to be conducted at the unscheduled visit depend on the reason for the visit. POE and ADA analyses should only be performed at unscheduled visits that are conducted for safety reasons when safety labs are collected for the management/monitoring of an AE. When a series of unscheduled visits is needed for the monitoring of the same AE, the POE and ADA collection is not required if already done at the first unscheduled visit of the series. Additional collection of samples for POE and ADA analysis should be performed per Investigator's judgment.
- d) PP NRS to be recorded by subjects once daily in the evening. SD NRS to be recorded by subjects once daily in the morning and if possible, within 1 hour of getting out of bed.
- e) Patient-reported outcome assessments and designated safety measurements (including AE and concomitant therapies/procedures assessments) should occur before Investigator assessments, laboratory sample collections, and study drug administration.
- Subjects with a history of asthma will complete the ACT testing at all visits. Subjects with a new (de novo) diagnosis of asthma will complete the ACT testing beginning from de novo diagnosis and at all subsequent scheduled visits.

Statistical Analysis Plan for Interventional Studies


g) Respiratory exams and PEF measurements are required at these visits for subjects with a medical history of asthma or newly-diagnosed (de novo) asthma only. Whenever possible, it is preferable that the PEF measurements be performed before noon or at the same time during each study visit. Subjects should be asked to withhold asthma medication on study

visit days until after PEF testing is complete, to the extent it does not pose an undue risk to the subject.

h) Vital signs will include pulse rate, systolic and diastolic blood pressure (after the subject has been sitting for at least 5

minutes), and body temperature.

i) 12-lead ECGs should be performed in the supine position and before any scheduled vital sign measurements and blood

draws.

j) Subjects should be reminded to be well hydrated and fast for at least 8 hours before the visit(s) when clinical chemistry

testing is planned. See Section 12.5 of the protocol for details.

k) Only for females of childbearing potential. If UPT is positive, it must be confirmed with a serum pregnancy test. Pregnancy

test results must be available prior to the administration of the study drug.

For postmenopausal subjects (i.e., no menses for 12 consecutive months), confirm status with a high FSH level in the postmenopausal range unless previously confirmed as part of a lead-in study. The blood chemistry sample at the baseline

visit (V1) will also be used for an FSH test for the confirmation of postmenopausal status, if applicable.

m) At scheduled visits with laboratory, POE, and/or ADA assessments, the samples are to be collected before study drug

injection(s). As a guideline, POE and ADA samples should be collected at approximately the same time of day throughout

the study, to the extent possible.

n) Study drug reconstitution will be performed by the pharmacist (or other qualified personnel), and complete reconstitution

confirmed, prior to delivery for injection.

o) Clinic staff will provide injection training (or re-training, as needed) for subjects willing and able to self-inject study drug.

Subjects will then be allowed to inject study drug. Based on the subject's preference, clinic staff can also perform all

injections.

p) After study drug administration, subjects should be monitored closely for any signs or symptoms of hypersensitivity reaction

before being discharged.

q) If a study visit occurs outside of the visit window, study drug injection(s) can still be administered provided there is a minimum of 3 weeks but not more than 5 weeks since the last injection. If 5 weeks or more, the next study drug injection should then

occur at the next planned visit. Future visits should be scheduled as soon as possible and within the required windows

based on the baseline/Day 1 visit date, while maintaining the minimum 3-week interval between doses.

The dose will depend on the dose received in the LTE lead-in study RD.06.SPR.202699.

## 5. Endpoints

### 5.1. Primary Efficacy Endpoints

Time from baseline to relapse, defined as meeting at least 1 of the following criteria:

- Increase in (weekly average of the) PP NRS score ≥4 points from baseline
- Increase in IGA score ≥2 points from baseline

## 5.2. Secondary Efficacy Endpoints

The secondary efficacy endpoints are as follows:

- Proportion of subjects with increase in PP NRS score ≥4 points from baseline at each scheduled visit
- Proportion of subjects maintaining IGA success, defined as IGA score of 0 (clear) or 1 (almost clear) at each scheduled visit
- Proportion of subjects with increase in IGA ≥2 points from baseline at each scheduled visit
- Absolute and percent change from baseline in PP NRS at each scheduled visit
- Absolute and percent change from baseline in Sleep Disturbance Numeric Rating Scale (SD NRS) at each scheduled visit
- Change from baseline in DLQI at Week 16 and Week 24

## 5.3. Safety Endpoints

The safety endpoints of this study are as follows:

- Incidence and severity of AEs, including treatment-emergent AEs (TEAEs), AESIs, serious AEs (SAEs), treatment-related AEs, and AEs that lead to discontinuation.
- Physical examination and Vital signs
- Clinical laboratory tests
- Electrocardiogram
- Peak expiratory flow
- Asthma Control Test (ACT)


- Anti-drug antibody (ADA) concentrations
- Incidence of positive ADA assays
- Nemolizumab (CD14152) serum concentrations

6. Analysis Sets

6.1. Intent-to-Treat Population

The intent-to-treat (ITT) population will consist of all randomized subjects. All primary and secondary

efficacy endpoints will be analyzed based on the ITT population. All analyses on the ITT population will be

analyzed under the treatment group "as randomized".

6.2. Safety Population

The safety population will comprise all randomized subjects who receive at least 1 dose of study drug. All

safety data will be summarized based on the safety population under the treatment group "as treated".

6.3. Proof of Exposure Analysis Population

The proof of exposure (POE) analysis population will include all subjects in the safety population who

provide at least 1 measurable post-baseline evaluable drug concentration value.

6.4. Per-Protocol Population

The Per-Protocol (PP) population will consist of all subjects in the ITT population who have no major

protocol deviations that would have a significant effect on the efficacy of the study treatment (see Section

6.5). Only primary and selected secondary endpoints will be analyzed using the Per-Protocol Population,

under the treatment group as randomized.

6.5. Protocol Deviations

Protocol deviations will be recorded by the Clinical Research Associate (CRA) in the Clinical Trial

Management System (CTMS). All protocol deviations will be categorized by the associated deviation type

and will be assessed individually on a regular basis on whether they are major or minor. Details can be

found in the Protocol Deviation and Non-compliance Management Plan.

Major protocol deviations that are analysis relevant lead to an exclusion of the subject from the per-protocol

population. A case by case decision regarding exclusions of subjects from the per-protocol analysis will be

made in a blind data review meeting (BDRM) which will take place prior to unblinding the study. The criteria

for exclusion from the Per-Protocol Population will be specified in the BDRM Preparation Plan. Only major

protocol deviation which have a significant effect on the efficacy will result in exclusion from the Per-Protocol

Population.

Individual deviations (major and minor) will be presented in a data listing on the ITT population. A

summary table for number and percentage of subjects with major protocol deviation will be generated by

type of deviation and treatment group for the ITT population.

Statistical Analysis Plan for Interventional Studies


Protocol deviations incurred as a direct result of the COVID-19 pandemic should be specifically recorded and presented as a COVID-19 deviation. The number and percentage of subjects with major (including COVID-19) deviation will be provided by type of deviation and treatment group for the ITT population.

All protocol deviations will be listed.

### 7. Estimands

The primary efficacy endpoints will be evaluated and assigned to treatment at the time of randomization based on ITT Population. The estimand is defined to address the scientific question relevant to subjects who are able to complete treatment with a response assessment without further medication being required, other than permitted medication.

An intercurrent event is an event which occurs after start of treatment and thus complicates the description and interpretation of treatment effects. Table 7-1 below lists potential intercurrent events and the strategy to deal with them for the estimand. The estimands for endpoints are defined in

Table 7-2

Table 7-1: List of Intercurrent Events

| Intercurrent Event | Strategy to Deal With<br>Intercurrent Event Within<br>Analysis | Assessment of Subject |
|---|---|---|
| Treatment discontinuation | While on Treatment Strategy | Any data collected after a treatment discontinuation will be censored |
| Use of prohibited medication | While on treatment strategy | Any data collected after a use of prohibited medication will be censored |

Table 7-2: Estimands for primary Endpoint

| Endpoints | Estimands |
|---|---|
| Time to relapse meeting | Treatment: randomized treatment with subcutaneous injections of |
| at least 1 of the defined criteria* | nemolizumab or placebo at Week 0, 4, 8, 12, 16, and 20 |
| Ciliena | Population: ITT population |
| | Endpoint: Time to relapse meeting at least 1 of the defined criteria |
| | Intercurrent events: Time to relapse will be censored at the last |
| | observation prior to treatment discontinuation or use of prohibited |
| | medication |


| Endpoints | Estimands |
|-----------|----------------------------------------------------------|
| | Summary measure: Hazard ratio of nemolizumab and placebo |

<sup>\*</sup>the time to relapse which is defined as meeting at least 1 of the following criteria:

- Increase in (weekly average of the) PP NRS score ≥4 points from baseline
- Increase in IGA score ≥2 points from baseline

8. General Aspects for Statistical Analysis

8.1. General Methods

• All data will be listed, and summary tables will be provided.

• Unless otherwise specified, summaries will be presented for each treatment, if indicated, by visit.

• Continuous variables will be summarized using the number of observations (n), mean, standard

deviation (SD), median, minimum and maximum. Categorical variables will be summarized using

number of observations (n), frequency and percentages of subjects

• Unless otherwise stated, all statistical tests will be two-sided and conducted at the 5% level; all

presented confidence intervals (CIs) will be two-sided 95% CIs.

8.2. Key Definitions

The 24-week treatment period is defined as Day 1/Baseline to Week 24. If early discontinued during

treatment period, it is defined as the period until 4 weeks (<=28 days) after last dosing date or early

termination date whichever is earlier.

The Baseline value is defined as the last non-missing value before the first dose of study drug. In case

that the date of first injection is not available, the date of randomization is considered.

For diary data (PP NRS, SD NRS), the Baseline values will be week 52 value from LTE trial.

The date of first treatment is defined as the date of first injection of study drug.

The date of last treatment is defined as the date of last injection of study drug.

Study day is defined as the number of days from the date of first treatment (randomization date if not

treated) and will be calculated as follows:

• If the event date ≥ date of first treatment, then study day = event date – date of first treatment + 1.

Treatment Day 1 is therefore defined as the day of first treatment.

If the event date < date of first treatment, then study day = event date - date of first treatment.</li>

• If subject is randomized, but not treated, then study day = event date - date of randomization.

A subject's date of last participation in the trial is the last date of contact.

Only the subjects infected by COVID-19 during study participation will be considered subjects with

COVID-19 infection.

Statistical Analysis Plan for Interventional Studies


8.3. Missing Data

When analyses are not based on OC, the primary method to impute the missing values will be as follows:

Continuous Endpoints: For continuous secondary endpoints during treatment period, the MMRM

approach will be used to handle the missing data.

Binary Endpoints: For binary secondary endpoints during treatment period, missing data will be imputed

to failure.

Adverse events and concomitant medications/procedures: Missing assessment times will have

imputed times for the purposes of assessing treatment emergence for AEs or classifying

medications/procedures into prior/concomitant. However, the assessment date and time (start date, stop

date, and time if collected from CRF) without imputation will be presented in the listings.

For the start of a concomitant medication/procedure or AE:

• Only the year is reported: If the subject received the first study drug dose in the year reported, then

the date of the first dose of study drug will be used as the start date; otherwise, January 1 of the

year reported will be used as the start date.

• The month and year are reported: If the subject received the first study drug in the month and year

reported, then the date of the first dose of study drug will be used as the start date; otherwise, the

first day of the month and year will be used as the start date.

The time is collected but missing: If the start date is the same as the date the subject started

receiving study drug, then the time of the first dose of study drug will be used as the start time;

otherwise, 00:00 will be used as the start time.

For the end of a concomitant medication/procedure or AE:

• Only the year is reported: The earlier between December 31 of the year reported and the date of

the last study contact with the subject will be used as the stop date.

The month and year are reported: The earlier between the last date of the month and year reported

and the date of the final contact with the subject will be used as the stop date.

The time is collected but missing: 23:59 (or 23:59:59 if collected up to seconds) will be used as the

stop time.

If an AE has the start date completely missing and the stop date on/after the first dose date of study drug, this AE will be considered as treatment emergent (TEAE).

If a medication/procedure has the stop date completely missing, this medication/procedure will be considered as ongoing and concomitant. If the start date of a medication/procedure is completely missing and impossible to identify different by stop date, this medication will be considered as concomitant.

#### 8.4. Visit Windows

Efficacy by-visit summaries will use the analysis visit. All visits including unscheduled and early termination visits will be windowed based on the analysis visit window in Table 8-1 which is based on study day. If multiple measurements are taken within the same window, the one taken closest to the target study day will be used for the analysis. If there are multiple measurements with same difference from target day, the later assessment should be used for the analysis.

Table 8-1: Analysis Visit Window

| Analysis Visit | Target Study Day | Visit Window (IGA) | Visit Window (DLQI) |
|---|---|---|---|
| Baseline | 1 | ≤ 1 | ≤ 1 |
| Week 4 | 29 | 2 to 42 | N/A |
| Week 8 | 57 | 43 to 70 | N/A |
| Week 12 | 85 | 71 to 98 | N/A |
| Week 16 | 113 | 99 to 126 | 2 to 140 |
| Week 20 | 141 | 127 to 154 | N/A |
| Week 24 | 169 | 155 to 210 | 141 to 210 |
| Week 32 Follow-up | 225 | >211 | N/A |

All daily diary efficacy data will be classified into analysis visits as described in Table 8-2 considering the data during the 7 days immediately preceding the target day of analysis visit.

Analysis visit of diary (ePRO) data will be defined depending on the data collection as below.

#### Consecutive daily assessment:

For the evening assessments (PP NRS), the daily data collected up to Week 24 will be classified into analysis visits considering the data during the 7 days immediately preceding the target study day of analysis visit. Similarly, for the morning assessment (SD NRS, morning sleep diary), the 7 days data up to the target study day will be classified into analysis visit. Details of the analysis visit window are in Table 8-2 below.

Table 8-2: Analysis Visit Window for Evening and Morning Assessments

| Analysis Visit | Target Study Day | Visit Window for evening | Visit Window for morning |
|---|---|---|---|
| | of Analysis Visit | assessment (PP NRS, AP | assessment (SD NRS, |
| | | NRS) | morning sleep diary) |
| Baseline | 1 | -7 to -1 | -6 to 1 |
| Week 1 | 8 | 1 to 7 | 2 to 8 |
| Week 2 | 15 | 8 to 14 | 9 to 15 |
| Week 3 | 22 | 15 to 21 | 16 to 22 |
| Week 4 | 29 | 22 to 28 | 23 to 29 |
| Week 5 | 36 | 29 to 35 | 30 to 36 |
| Week 6 | 43 | 36 to 42 | 37 to 43 |
| Week 7 | 50 | 43 to 49 | 44 to 50 |
| Week 8 | 57 | 50 to 56 | 51 to 57 |
| Week 9 | 64 | 57 to 63 | 58 to 64 |
| Week 10 | 71 | 64 to 70 | 65 to 71 |
| Week 11 | 78 | 71 to 77 | 72 to 78 |
| Week 12 | 85 | 78 to 84 | 79 to 85 |
| Week 13 | 92 | 85 to 91 | 86 to 92 |
| Week 14 | 99 | 92 to 98 | 93 to 99 |
| Week 15 | 106 | 99 to 105 | 100 to 106 |
| Week 16 | 113 | 106 to 112 | 107 to 113 |
| Week 17 | 120 | 113 to 119 | 114 to 120 |
| Week 18 | 127 | 120 to 126 | 121 to 127 |
| Week 19 | 134 | 127 to 133 | 128 to 134 |
| Week 20 | 141 | 134 to 140 | 135 to 141 |
| Week 21 | 148 | 141 to 147 | 142 to 148 |
| Week 22 | 155 | 148 to 154 | 149 to 155 |
| Week 23 | 162 | 155 to 161 | 156 to 162 |
| Week 24 <sup>a</sup> | 169 | 162 to 175 | 163 to 176 |
| Early | UN | 7 days prior until Early | 6 days prior until early |
| Termination* | | termination visit (excluding | termination visit (including |
| | | early termination visit date) | early termination visit date) |

<sup>&</sup>lt;sup>a</sup> First 7 days data available will be used for weekly average calculation.

<sup>\*</sup>For subjects with early termination, if weekly average is not available based on the slotting, additional analysis window was added and will be assigned to the week based on the slotting above. i.e., if subject


early terminated day 142, and week 21 is not available, the new window defined will be used to determine the weekly average at that week.

Safety and pharmacokinetics data will not be windowed for by-visit summary. i.e., scheduled visit data will be used for analysis.

### 8.5. Subgroups

Subgroup analysis will not be conducted in this study, regarding the small sample size.


9. Demographic, Other Baseline Characteristics and Medication

9.1. Subject Disposition and Withdrawals

All subjects of the ITT population will be accounted for in this study.

Subject accounting will summarize subjects randomized and randomized but not treated for all subjects by

overall and site.

Subject accounting by visit will be summarized by treatment group and overall at each visit (scheduled visits

only).

Subject disposition will be summarized based on the ITT population by treatment and overall. Summaries

will include subjects randomized, subjects randomized but not treated, subjects treated, subjects completed

treatment, subjects discontinued treatment, primary reason for discontinuation of treatment (including

summary of subjects who stopped treatment due to COVID-19), subjects completed the study, subjects

discontinued from the study, primary reason for discontinuation from the study (including summary of

subjects who discontinued due to COVID-19) and subjects completed Follow-up. Subjects who stopped

treatment or discontinued study due to COVID-19 will be identified using other specify field in CRF.

Subject disposition will also be summarized by site on the ITT population.

Subjects in each analysis population (ITT, SAF, PP, POE analysis population) will be summarized by

treatment group on the ITT population.

In addition, time (days since the first dose of study drug) to permanent discontinuation of study drug by

reason for discontinuation will be displayed graphically in subjects having permanently discontinued from

the study drug.

Randomization, study completion, drug completion, visit dates will be listed for the ITT population.

Additional listings of discontinuation reason, missed visit and missed assessment for subjects who

discontinued due to COVID-19 will be presented for the ITT population.

Analysis populations will be summarized and listed on the ITT population.

9.2. Demographic and Baseline Disease Characteristics

Summary statistics for demographic and other Baseline disease characteristics will be presented for the

ITT, SAF, PP and POE analysis population.

Age (years), height (cm), weight (kg), and BMI (kg/m²) will be summarized using summary statistics for

continuous variables. Age groups (18-65, and > 65), sex, region (Europe, North America, and Asia Pacific),

race, ethnicity, and smoking history will be summarized using the summary statistics for categorical

variables. Weight will additionally be presented for each subgroup < 90 kg and ≥ 90 kg as well as dosing

regimen (1 or 2 injections).

The Baseline disease characteristics IGA, weekly average PP NRS, weekly SD NRS and baseline DLQI

will be summarized. IGA, will be summarized as a categorical variable.

A summary table for the stratification factor dosing regimen will be provided to show any discrepancies

between what was reported through Interactive Voice Response System (IVRS)/Interactive Web Response

System (IWRS) versus eCRF data (at baseline visit).

All demographic and baseline disease characteristics data will be listed on the ITT population.

9.3. **Medical History** 

Medical history will be collected only at baseline and will be coded using Medical Dictionary for Regulatory

Activities (MedDRA, Version 25.0).

Medical history will be summarized by treatment group. The summary will include number and percentage

of subjects reporting each system organ class (SOC) and preferred term (PT) and will be sorted

alphabetically by SOC and descending frequency of PT within SOC in the Nemolizumab treatment group.

Summary tables will be presented for the ITT population.

Medical history data listings will be presented by subject number, start date, stop date, SOC, and PT for

the ITT population.

9.4. **Medical and Surgical Procedure** 

Medical and surgical procedures will be coded using the latest version of Medical Dictionary of Regulatory

Activities (MedDRA).

Prior medical and surgical procedures are defined as those which have been stopped before first treatment.

Concomitant medical and surgical procedures will be defined as those started or stopped on or after the

first treatment, or were ongoing during the study. If a procedure is started before the first treatment but is

ongoing or stopped on or after the first treatment, it will be considered concomitant.

Procedures during treatment period will be defined from start of treatment till 4 weeks (<= 28</li>

days) after the last treatment or early discontinuation date whichever is earlier.

Procedures during follow-up period is defined from post treatment period (4 weeks (> 28 days)

after the last treatment or early discontinuation date, whichever is earlier) to follow-up visit date.


If the stop date and 'ongoing' are missing then the procedure will be considered concomitant. If stop date

is partially missing, the procedure will be considered concomitant unless the non-missing part of date

proves it ended prior to the first treatment date.

The following medical and surgical procedures (prior and concomitant) will be summarized by treatment

group using the number and percent of subjects reporting each SOC and PT and sorted alphabetically by

SOC and descending frequency of PT within SOC in the Nemolizumab treatment group. Summary tables

will be presented for the ITT population.

Prior procedure

Concomitant procedure during treatment period

Concomitant procedure during follow-up period

Medical and surgical procedures listings will be presented by treatment group on the ITT population and

sorted by subject number, start date, stop date, SOC, and PT.

Medication 9.5.

Medications will be classified and summarized on the ITT population as follows:

Prior medications are defined as those which stop before the first injection of study drug during the study.

Concomitant medications are defined as those started, stopped or ongoing on or after the first injection of

study drug.

Medication during treatment period is defined from start of treatment till 4 weeks (<= 28 days) after

the last treatment or early discontinuation date whichever is earlier.

Medication during follow-up period is defined from post treatment period (4 weeks (> 28 days) after

the last treatment or early discontinuation date, whichever is earlier) to follow-up visit date.

If the stop date and 'ongoing' are missing then the medication will be considered as concomitant medication. If stop date is partially missing, the medication will be considered as concomitant unless the non-missing

part of date proves it ended prior to the first treatment date.

Medications (prior, concomitant and prohibited medications) will be coded using Version B3 Sep2021 of

the World Health Organization's Drug Dictionary (WHO DD). Preferred Anatomical Therapeutic Chemical

(ATC) coding will be performed.

The following summaries by ATC level 2, ATC level 4 and preferred term (PT) will be produced on the ITT

population. Subjects with more than one medication in a given ATC level and preferred name will be

counted only once in that category. It will be sorted ATC level alphabetically and descending frequency in

PT within ATC level term.


• Prior medication

Concomitant medication during treatment period

Concomitant medication during follow-up period

Prohibited medication during treatment period

Prohibited medication during follow-up period

All medications (prior and concomitant medications, prohibited medications) will be listed for the ITT

population.

9.6. Extent of Exposure

Following parameters will be summarized:

• Treatment duration (in days) is calculated as follows, where date of first treatment is defined as the

first day: [(date of last treatment - date of first treatment) + 1].

Total dose administered (mg) will be calculated as the sum of all doses of study drug administered.

• Total dose planned (mg) will be calculated as the sum of all doses of study drug planned

(dispensed) according to the treatment schedule of the treatment group.

The number of subjects who missed at least one dose

The number of subjects who missed at least one dose due to COVID-19

The number of doses missed

The number of doses missed due to COVID-19

Note: The missed dose due to COVID-19 are captured as other-reason reported in CRF.

9.7. Treatment Compliance

Treatment compliance will be assessed through the treatment records and drug dispensation logs. As study

drug is administered in the clinic, treatment compliance will be overseen and documented by the

investigator and study staff (using the treatment records and drug accountability records).

Treatment compliance (%) is calculated as the total number of actual injections / the total number of

expected injections \* 100. The total number of actual injections is counted based on collected study drug

administration data. The total number of expected injections is counted based on the dosage schedule and

dispensed as per protocol.

## 10. Efficacy

Unless otherwise stated, all efficacy analyses will be performed on the ITT population.

All efficacy variables will be summarized by treatment group at each analysis visit. The primary comparison of interest is Nemolizumab compared to placebo.

#### 10.1. Primary Efficacy Endpoints

### 10.1.1. Primary Analysis of Primary Efficacy Endpoint

The primary endpoint is the time to relapse which is defined as meeting at least 1 of the following criteria:

- Increase in (weekly average of the) PP NRS score ≥4 points from baseline
- Increase in IGA score ≥2 points from baseline;

For primary endpoint, any subjects with missing data for PP NRS and IGA Score both at visit will be censored at the respective timepoint. If any one of PP NRS or IGA Score data is available for the visit, calculation for primary endpoint will be made using available results. If a subject has taken prohibited medication at any point of time during treatment period, then subject will be censored at the respective visit.

The primary endpoint will be analyzed using Cox proportional hazard model with treatment group, dosing regimen as a factor, and baseline PP NRS score and IGA score as covariates on ITT population. The estimated hazard ratio and the corresponding 95% CI will be presented. A supportive analysis also will be performed using Per-Protocol Population.

Kaplan-Meier survival plots will also be presented for time to relapse. The median time, 25<sup>th</sup> and 75<sup>th</sup> quantiles along with corresponding CI will be presented using ITT/PP.

Censoring rule for primary endpoint variable is as follows:

| Situation | Date of Progression or Censoring | Outcome |
|---|---|---|
| Relapse as described | Date of Relapse | Event |
| Subject withdrawn without relapse | Date of last efficacy assessment (PP NRS and IGA) prior to withdrawal | Censored |
| Treatment Discontinuation | Date of last efficacy assessment (PP NRS and IGA) prior to Treatment Discontinuation | Censored |
| Prohibited medication without relapse | Date of last efficacy assessment (PP NRS and IGA) prior to prohibited medication | Censored |
| Completes the study without relapse | Date of Week 24 completion | Censored |
| No Efficacy assessment | Date of study Day 1 | Censored |

## 10.1.2. Sensitivity Analyses of Primary Efficacy Endpoint

Sensitivity analyses for primary endpoint will be conducted in order to test for the robustness of the primary analyses. The following sensitivity analyses will be conducted:

- Same analysis on Per-Protocol Population as mentioned in 10.1.1.
- 'Actual strata of randomization' instead of 'stratum at the randomization' for subjects stratified incorrectly.
- Removal of COVID-19 affected visits (i.e. exclusion of subjects from visit, if visit was missed due to COVID-19.) This is analysis will be performed only if >2% subjects have missing data due to COVID-19.

## 10.2. Secondary Efficacy Endpoints

The following secondary endpoints are to be analysed at the scheduled visits:

| Endpoint | Analysis Visit | | Analysis to be done | Statistical | |
|---|---|---|---|---|---|
| | | | | on which Population | Tests |
| Proportion of subjects maintaining IGA | Baseline, | Week | 4, | On the ITT and Per- | CMH |
| success at each scheduled visit | Week 8, | Week | 12, | Protocol Population | |
| | Week 16, | Week | 20, | | |
| | Week 24 | | | | |
| Proportion of subjects with increase in | Baseline, | Week | 4, | On the ITT and Per- | CMH |
| IGA ≥2 points from baseline at each | Week 8, | Week | 12, | Protocol Population | |
| scheduled visit | Week 16 | | | | |
| Proportion of subjects with increase in | Baseline, | Week | 4, | On the ITT and Per- | CMH |
| PP NRS score ≥4 points from baseline | Week 8, | Week | 12, | Protocol Population | |
| at each scheduled visit | Week 16, | Week | 20, | | |
| | Week 24 | | | | |
| Absolute and percent change from | Baseline, | Week | 4, | On the ITT and Per- | ANCOVA |
| baseline in PP NRS at each scheduled | Week 8, | Week | 12, | Protocol Population | |
| visit | Week 16, | Week | 20, | | |
| | Week 24 | | | | |
| Absolute and percent change from | Baseline, | Week | 4, | On the ITT | MMRM |
| baseline in PP NRS at each scheduled | Week 8, | Week | 12, | | |
| visit | Week 16, | Week | 20, | | |
| | Week 24 | | | | |

| Endpoint | Analysis Visit | Analysis to be done | Statistical |
|---|---|---|---|
| | | on which Population | Tests |
| Absolute and percent change from | Baseline, Week 4, | On the ITT and Per- | ANCOVA |
| baseline in SD NRS at each scheduled | Week 8, Week 12, | Protocol Population | |
| visit | Week 16, Week 20, | | |
| | Week 24 | | |
| Absolute and percent change from | Baseline, Week 4, | On the ITT | MMRM |
| baseline in SD NRS at each scheduled | Week 8, Week 12, | | |
| visit | Week 16, Week 20, | | |
| | Week 24 | | |
| Change from baseline in DLQI at each | Baseline, Week 16, | On the ITT Population | ANCOVA |
| visit | Week 24 | | |

Abbreviations: CMH= Cochran-Mantel-Haenszel; DLQI=Dermatology Life Quality Index; IGA=Investigator Global Assessment; PP=Peak Pruritus; SD=Sleep Disturbance.

Binary secondary efficacy endpoints will be analyzed using a Cochran-Mantel-Haenszel test adjusted for dosing regimen based on OC and imputation with missing efficacy response considered as the non-responder (i.e., IGA success) and missing relapse response considered as a relapse (i.e., increase in PP NRS or IGA). The estimate of treatment unadjusted and strata-adjusted differences with the corresponding two-sided 95% confidence intervals, and p-values from the CMH test will be presented.

Continuous secondary endpoints will be analyzed using analysis of covariance (ANCOVA) based on OC with treatment group and dose regimen as factors, and baseline value as the covariate. In addition, for PPNRS and SDNRS endpoints, the mixed effect model for repeated measure (MMRM) approach based analysis will be repeated on OC, including treatment group and dose regimen as factor, visit, interaction term between treatment and visit along with corresponding baseline value as independent covariate. Kenward-Roger approximation is used to estimate denominator degrees of freedom. An unstructured covariance is used to model the within-patient errors in the analysis. While applying the model, if convergence criteria not met with unstructured covariance matrix, then "Type = CS or type =ar(1)" covariance matrix will be applied to achieve convergence of the model. The matrix with the minimum AIC criteria will be selected for the further analysis. For both analyses, the least squares means, estimated standard error, and 95% confidence interval (CI) for each endpoint will be presented for each treatment group and analysis visit; the estimated treatment difference for each endpoint at each analysis visit will be summarized by presenting the difference in least squares means between treatment groups, the two-sided 95% CI, and associated p-value as well.

All secondary endpoints will be presented descriptively using OC.

#### 10.2.1. Investigator's Global Assessment (IGA)

The IGA is a 5-point scale used by the Investigator or trained designee to evaluate the global severity of PN and the clinical response to a treatment (see Table 10-1).

Table 10-1: Investigator Global Assessment Scale

| 0 | Clear | No nodules |
|---|--------------|---------------------------------------|
| 1 | Almost Clear | Rare palpable pruriginous nodules |
| 2 | Mild | Few palpable pruriginous nodules |
| 3 | Moderate | Many palpable pruriginous nodules |
| 4 | Severe | Abundant palpable pruriginous nodules |

IGA treatment success is defined as 0 (clear) or 1 (almost clear) on the IGA scale.

IGA will be collected at Baseline/Day 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and Early Termination or any unscheduled visit. In case of missing assessment at Baseline, the last available assessment prior study drug administration will be considered as Baseline.

IGA will be summarized as a categorical and continuous variable at each analysis visit. Absolute change from Baseline for the IGA score will also be presented in the summary on the ITT and Per-Protocol Population.

The proportion of subjects maintaining IGA success and subjects with increase in IGA  $\geq$  2 points from baseline will be summarized on the ITT based on OC. The estimate of treatment unadjusted and strata-adjusted differences with the corresponding two-sided 95% confidence intervals, and p-values from the CMH test will be presented.

The analysis will be repeated:

- on Per-Protocol Population, based on OC
- on ITT population, imputing missing values with non-responder imputation

Line plot for proportion of subjects maintaining IGA success and proportion of subjects with increase in IGA ≥ 2 points from baseline, both using non-responder imputation, will be for the ITT Population.

### 10.2.2. Pruritus Numeric Rating Scale (NRS)

The Pruritus NRS is a scale to be used by the subjects to report the intensity of their pruritus (itch) during the last 24 hours. Peak pruritus (PP NRS) is an assessment of the maximum itch intensity in that period.

Subjects will be asked the following question:



The Baseline PP NRS will be the score of Week 52 visit from LTE trial.

PP NRS at all follow-up visits will be determined as an average of 7 consecutive days data up to the target study day and will be set to missing if less than 4 days data are available. Subjects will receive instructions on how to record their PP NRS scores and will complete the assessment once daily in the evening throughout the clinical study (including the run-in and the follow-up period).

PP NRS will be determined by an average as described above at every week from Baseline to Week 24 as a continuous variable.

Descriptive summary of PP NRS (OC) will be provided on the ITT and Per-Protocol Populations. Absolute change and percent change from Baseline for the PP NRS will also be included in the summary on the ITT and Per-Protocol Populations.

Absolute change from Baseline in PP NRS will be analyzed using ANCOVA based on OC, including treatment group dose regimen as factors with baseline value as covariate. The least squares means (LSMeans), standard error of LSMeans, and 95% CI for change from baseline, as well as the difference in LSMeans between the treatment groups, the two-sided 95% CI, and associated p-value will be presented. Percentage change from Baseline in PP NRS will not be analyzed because of the small sample size and potential high skewness of the data.

The analysis will be repeated:

on Per-Protocol Population, based on OC

on ITT population, based on OC and using MMRM approach, including treatment group and dose regimen as factor, visit, interaction term between treatment and visit, and baseline value as covariate. Kenward-Roger approximation is used to estimate denominator degrees of freedom. An unstructured covariance is used to model the within-patient errors in the analysis. While applying the model, if convergence criteria not met with unstructured covariance matrix, then below mentioned covariance matrix will be applied to achieve convergence of the model. The matrix with the minimum AIC criteria will be selected for the further analysis.

- Compound Symmetry (CS)
- Ar(1) Autoregressive (1)

The proportion of subjects with PP NRS with  $\geq 4$  in increase from baseline will be summarized on the ITT based on OC. The estimate of treatment unadjusted and strata-adjusted proportion differences with the corresponding two-sided, 95% CI, and p-values from the CMH test will be presented. The analysis will be repeated:


- on Per-Protocol Population, based on OC
- on ITT population, imputing missing values with non-responder imputation

Line plot for proportion of subjects with PP NRS ≥ 4 increase will be presented on the ITT Population using non-responder imputation.

#### 10.2.3. Sleep Disturbance Numeric Rating Scale (SD NRS)

The SD NRS is a scale to be used by the subjects to report the degree of their sleep loss related to PN.

The baseline SD NRS will be the score of Week 52 visit from LTE trial.

Subjects will be asked the following question:



Descriptive summary of SD NRS (OC) will be provided on the ITT and Per-Protocol Population. Absolute change and percent change from Baseline will also be included in the summary.

Absolute change from Baseline in SD NRS will be analyzed using ANCOVA based on OC, including treatment group dose regimen as factors with baseline value as covariate. The least squares means (LSMeans), standard error of LSMeans, and 95% CI for change from baseline, as well as the difference in LSMeans between the treatment groups, the two-sided 95% CI, and associated p-value will be presented. Percentage change from Baseline in SD NRS will not be analyzed because of the small sample size and potential high skewness of the data.

The analysis will be repeated:

on Per-Protocol Population, based on OC

on ITT population, based on OC and using MMRM approach, including treatment group and dose regimen as factor, visit, interaction term between treatment and visit, and baseline value as covariate. Kenward-Roger approximation is used to estimate denominator degrees of freedom. An unstructured covariance is used to model the within-patient errors in the analysis. While applying the model, if convergence criteria not met with unstructured covariance matrix, then below mentioned covariance matrix will be applied to achieve convergence of the model. The matrix with the minimum AIC criteria will be selected for the further analysis.

- Compound Symmetry (CS)
- Ar(1) Autoregressive (1)

\_


10.2.4. Dermatology Life Quality Index

The DLQI is a validated 10-item questionnaire covering domains including symptoms/feelings, daily

activities, leisure, work/school, personal relationships, and treatment.

The subject will rate each question ranging from 0 (not at all) to 3 (very much). The DLQI total score is

calculated by summing each questionnaire. Total score will have a maximum score of 30 and a minimum

of 0. The higher score indicated a poorer quality of life.

DLQI will be collected at Baseline, Week 16, Week 24 and Early Termination. DLQI total score will be

summarized as a continuous variable using OC on the ITT Population. Absolute change and percentage

change from Baseline in DLQI total score will also be summarized.

Absolute change from Baseline in DLQI will be analyzed using ANCOVA based on OC, including treatment

group dose regimen as factors with baseline value as covariate. The least squares means (LSMeans),

standard error of LSMeans, and 95% CI for change from baseline, as well as the difference in LSMeans

between the treatment groups, the two-sided 95% CI, and associated p-value will be presented. Percentage

change from Baseline in DLQI will not be analyzed because of the small sample size and potential high

skewness of the data.

## 11. Pharmacokinetics

The serum concentration of Nemolizumab will be assessed at Baseline, Week 24 and Early Termination visit. PK analyses are required during any unscheduled visit conducted for safety reasons. As a guideline, PK samples should be collected at approximately the same time of day throughout the study, to the extent possible, before study drug injection (pre-dose samples).

#### 11.1. Pharmacokinetic Concentration Presentation

Serum concentration data (unit: ng/mL) will be summarized on the POE analysis population by visit and by dosing regimen from Baseline and Week 24, using the following statistics: arithmetic mean, SD, coefficient of variation (CV), geometric mean, geometric CV, median, minimum, maximum, 95% CI of the arithmetic mean, and number below the limit of quantification (BLQ).

Mean and individual (spaghetti plot) serum concentration(s) will be plotted by visit and by dosing regimen on both a linear and semi-logarithmic scale on the POE analysis population (2 plots).

Individual serum concentrations will be listed on the POE analysis population.

12. Immunogenicity

Blood samples to assess anti-Nemolizumab ADA will be collected at Baseline, Week 24 and Early

Termination. Immunogenicity analyses will be summarized on the POE analysis population.

Details related to the processing of serum samples and the assessments of ADA will be described in the

bioanalytical plan, which will be finalized before the beginning of sample analysis. Results will be described

in the bioanalytical report, which will be included as an appendix in the final clinical study report.

Incidence of positive ADA results will be summarized (absolute occurrence and percent of subjects) and

plotted by dosing regimen at each visit. The concentration of ADA titer (ng/mL) and neutralizing antibodies

(ng/mL) will be summarized as continuous variables.

The number and percentage of subjects with treatment related ADA will be summarized by visit and dosing

regimen. A treatment-related ADA is defined when the Baseline or confirmatory ADA result is negative and

the post-baseline confirmatory ADA result is positive in the Nemolizumab treated group only.

Individual trough serum drug concentrations will be plotted over time in ADA-positive versus ADA-negative

subjects.


13. Safety

All safety data will be summarized and listed on the SAF population.

Safety assessments will be conducted for all subjects at the baseline visit and at every subsequent visit.

Safety will be assessed on the basis of AEs (including TEAEs, AESIs, and SAEs), physical examination

and vital signs, clinical laboratory tests, electrocardiogram (ECG) and respiratory assessments. Summary

of all safety endpoints will be presented for each treatment group.

13.1. Adverse Events

AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA) Version 24.1.

Treatment-emergent AEs (TEAEs), defined as those AEs occurring after the first administration of study

treatment until the end of the follow-up period, will be tabulated in frequency tables by System Organ Class

(SOC) and Preferred Term (PT) based on the MedDRA for treatment and follow-up periods. Missing date

information will be handled using the algorithm described in Section 8.3.

TEAEs during treatment period are defined as AEs with onset date on or after the first dose date till 4 weeks

after the last treatment or early discontinuation date whichever is earlier. TEAEs during follow-up period

are defined as AEs with onset date post treatment period (4 weeks after the last treatment or early

discontinuation date, whichever is earlier) to follow-up visit date.

AEs will be summarized using the number and percent of subjects reporting each SOC and PT and sorted

alphabetically by SOC and by descending frequency of PT within SOC.

Subjects who experienced multiple events within the same SOC will be counted once in the SOC summary.

Subjects who experienced multiple occurrences of events with the same PT will be counted once in the PT

summary.

When summarizing by causality or maximum severity, if a subject experiences more than 1 occurrence of

the same AE, the occurrence with the greatest severity and the closest association with the study drug will

be used in summary tables. TEAEs related to study drug/study procedure are those that are identified as

reasonable possibility. If relationship or severity are missing, the event will be considered as AE related to

study drug/study procedure or severe AE.

An AESI is a noteworthy treatment-emergent event for the study drug that should be monitored closely and

reported promptly. An AESI can be either serious or non-serious. Based on the potential risks of

Nemolizumab and the risks associated with biologics in general (i.e., class effects), the following AEs will

be considered as AESIs:

Injection-related reactions,

Newly diagnosed asthma or worsening of asthma,

- Infections
- COVID-19 infections
- Peripheral edema: limbs, bilateral,
- Facial edema
- Elevated ALT or AST (> 3 x ULN) in combination with elevated bilirubin (> 2 x ULN).

The following summary tables for TEAEs will be presented for all TEAEs (i.e., TEAE all causalities) and study drug related TEAEs separately by treatment period and follow-up period.

- Overall Summary of TEAEs :
  - Overall summary table includes summary of subjects reporting TEAEs,
  - TEAE by maximum severity [Mild, Moderate, Severe]
  - TEAE related to study drug,
  - o TEAE related to study drug by maximum severity [Mild, Moderate, Severe]
  - TEAE related to protocol procedure,
  - Serious TEAE,
  - Serious TEAE related to study drug,
  - TEAE of special interest,
  - TEAE leading to study drug interruption,
  - TEAE leading to study drug withdrawal,
  - TEAE leading to study discontinuation,
  - TEAE leading to death,
  - o TEAE related to study drug leading to death
- TEAEs by SOC and PT
- Serious TEAEs by SOC and PT
- TEAEs by SOC, PT and Maximum Severity
- Severe TEAEs by SOC and PT
- TEAEs leading to study drug withdrawal by SOC and PT
- TEAEs leading to study discontinuation by SOC and PT


TEAEs of special interest by category by SOC and PT

TEAEs occurred in >= 5% of subjects by SOC and PT

•

Adjudicated TEAEs by SOC and PT

TEAEs of Asthma and AESI reported by investigator with adjudication outcome by IAC

Confirmed adjudicated TEAEs by SOC, PT and maximum severity

TEAEs of special interest by category, SOC, PT and maximum severity

For overall study period which includes all periods (treatment and follow-up), the following summary tables will also be presented and repeated for all TEAEs (all causalities) and study drug related TEAEs.

Overall Summary of TEAEs

TEAEs by SOC and PT

For the subset of subjects with COVID-19 infection, the following summary tables will be provided additionally for all TEAEs and study drug related TEAEs, separately.

Overall summary of TEAEs

TEAEs by SOC and PT

Serious TEAEs by SOC and PT

TEAEs of Special Interest by category by SOC and PT

In addition, the exposure-adjusted incidence rate (i.e., number of subjects per 100 patient-years) will be summarized for all TEAEs (all causalities) and study drug related TEAEs during treatment period.

Exposure-adjusted incidence rates of TEAEs is defined as the number of subjects exposed to treatment and experiencing a certain event divided by the total time of all subjects who are at risk for the event. Specially, for subjects with no event the exposure time is the time from the first drug intake to the end of treatment period. Exposure years is calculated as last study drug exposure date minus first study drug exposure date plus one, divided by 365.25 which is the number of days count in a year. This exposure year calculated for each subject is then added cumulatively and is derived for each treatment arm. So each treatment arm will have one value for exposure years (also known as "patient years"). The exposure year calculation is different in case of subjects who have completed the study or discontinued from the study or having withdrawn from the study due to any reason. Only the event occurred during the treatment period will account for calculation.

Subject listings will be presented for all


TEAEs,

TEAEs of special interest,

Serious TEAEs,

Severe TEAEs.

TEAE leading to permanent discontinuation of study drug,

TEAEs leading to deaths.

Pre-treatment AE

13.2. Laboratory Evaluations

13.2.1. Clinical Laboratory Evaluations

The hematology laboratory analyses, clinical chemistry laboratory analyses, and urinalyses will be performed at a central laboratory. Reference ranges will be supplied by the central laboratory and used by the investigator to assess the laboratory data for clinical significance and pathological changes. Reference

ranges will be provided in the laboratory manual.

The following parameters will be reported for laboratory data.

• Hematology: Hemoglobin, hematocrit, white blood cell (WBC) count (with differential including

eosinophils), red blood cell (RBC) count, platelet count, and mean cell volume (MCV).

• Chemistry: Creatinine, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma

glutamyl transferase, alkaline phosphatase, lactate dehydrogenase, total bilirubin, direct bilirubin,

albumin, total protein, uric acid, sodium, potassium, calcium, chloride, glucose, urea, total cholesterol,

triglycerides, low-density lipoprotein, high-density lipoprotein, creatine phosphokinase (CPK). CPK

isoenzyme test will be performed only if CPK is elevated to >2.5 × upper limit of normal (ULN).

• Urinalysis: pH, glucose, ketones, blood, protein, leukocytes, nitrites, bilirubin, urobilinogen, and

specific gravity.

Laboratory assessments are performed at Baseline/Day 1, Week 12, Week 24, Early Termination and Week

32/Follow-up.

Hematology and chemistry laboratory data (absolute values and change from Baseline) will be summarized

as continuous variables by visit (Baseline and scheduled visits only). Urinalysis laboratory data will be

summarized by visit (Baseline and scheduled visits only). Last post-baseline, worst post-baseline and

maximum post-baseline results will also be included in the summaries and will include unscheduled visits


in the derivation. Worst post-baseline value will be defined as the highest or lowest value relative to the

reference range. Parameters will be presented in alphabetically order.

Shift tables will be generated using the reference ranges (Low, Normal, High and Missing) for hematology

and chemistry laboratory data. The number and percentage of subjects shifting from reference ranges

between Baseline and each visit (scheduled visits only) will be summarized. Last, worst and maximum post

baseline values will also be included in the shift tables and will include unscheduled visits in the derivation.

Summary of the number and percentage of subjects who met criteria of potential clinically significant (CS)

value will be summarized (scheduled visits only) for hematology, chemistry. Last, worst and maximum post-

baseline results will also be included in the summaries. Potentially CS ranges are listed in Section 20.2.

For statistical and graphical summaries of the laboratory tests, values below or above the limit of detection

(e.g. '< 3' or '> 500') are substituted with the lower limit of detection minus 1% for values below the lower

limit and are substituted with the upper limit of detection plus 1% for values above the upper limit (e.g. '< 3'

is substituted by '2.97', '> 500' is substituted by '505'). In data listings, the values are shown including the

< or > sign.

Distribution of continuous hematology and chemistry laboratory data (in particular, Aspartate

Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Total Bilirubin

(BILI), Creatinine Kinase (CK) and Leukocytes (WBC)) will be displayed graphically as boxplot by treatment

group for baseline and for each scheduled visits and the maximum post-Baseline (including unscheduled

visits in the derivation) values.

By-subject listing will be presented for all laboratory data. By-subject listing for subjects with at least one

abnormal result (out of reference range) will be provided for hematology and clinical chemistry. By-subject

listing for subjects with at least one potentially CS result will be provided for hematology, clinical chemistry.

All laboratory data will be listed for the Safety population.

13.2.2. Pregnancy Testing

All women of childbearing potential will have a serum pregnancy test at the baseline visit and urine

pregnancy tests (UPTs) at Baseline, Week 4, Week 8, Week 12, Week 16, Week 20 and Week 24, Early

Termination visit, and Week 32/Follow-up. Pregnancy test results must be available prior to the

administration of the study drug.

All confirmed pregnancy test results, premenses status and childbearing potential assessment results will

be listed on the Safety population.


13.2.3. Virology and TB Testing

Virology including hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C virus

(HCV), human immunodeficiency virus 1, and human immunodeficiency virus 2 antibodies may be

assessed at unscheduled visits for safety purposes based on Investigator judgment. Subjects with a positive

HBcAb and a negative HBsAg will also be assessed for hepatitis B surface antibody. Subjects with positive

HCV antibodies will have a confirmatory test for HCV (e.g., PCR). All virology results will be listed on the

Safety population.

Subjects may be assessed for active or latent tuberculosis (TB) at unscheduled visits for safety purposes

based on Investigator judgment. A subject who tests positive for latent TB (with a positive QuantiFERON-

TB Gold test) should be referred to the subject's treating physician for appropriate follow-up. All TB test

results will be listed on the Safety population.

13.3. Vital Signs

Vital signs will include pulse rate, systolic and diastolic blood pressure (after the subject has been sitting

for at least 5 minutes) and body temperature.

Vital signs will be collected at the at Baseline/Day 1, Week 4, Week 8, Week 12, Week 16, Week 20, and

Week 24, Early Termination visit, and at Week 32/Follow-up.

Height and weight will be measured at Baseline for all subjects. Weight assessments will be conducted at

Baseline/Day 1, and Week 24 and Early Termination.

All vital signs including height and weight (absolute values and change from Baseline) will be summarized

as continuous (Baseline and scheduled visits only). Last post-Baseline results (including unscheduled visits

in the derivation) will also be included.

The number and percentage of subjects who met criteria of potential CS value (Section 20.2) for vital signs

and weight will be summarized (Baseline and scheduled visits only). Last post-Baseline results (including

unscheduled visits in the derivation) will also be included.

Distribution of pulse rate, systolic and diastolic blood pressure will be displayed graphically as boxplot by

treatment group for Baseline and each scheduled visit and maximum post-Baseline (including unscheduled

visits in the derivation) values.

By-subject listing of subjects with potentially CS vital signs and weight will be provided.

All vital signs results will be listed on the Safety population.


13.4. ECG

A 12-lead electrocardiogram (ECG) will be performed and read centrally at Baseline/Day 1, Week 24 and

Early Termination visit.

All ECG data (absolute values and change from Baseline) will be summarized as continuous variables by

visit (Baseline and scheduled visits only). All parameters will be presented in alphabetically order.

The overall results of the ECGs recorded as 'Normal'. 'Abnormal, NCS' or 'Abnormal, CS' will be

summarized by treatment group and visit (scheduled visit only). Clinical significance will be determined by

the investigator.

Additionally, all ECG findings will be summarized with numbers and percentages by visit (Baseline and

scheduled visits only.

All ECG results will be listed on the Safety population.

13.5. Physical Examination

Following body system assessments will be performed at Baseline/Day 1, Week 12, Week 24, Early

Termination, and Week 32/Follow-up:

Head, ears, eyes, nose, throat, neck (including thyroid),

Skin/integumentary system (excluding PN),

· Cardiovascular system,

Respiratory system,

· Gastrointestinal system,

Musculoskeletal system,

Lymph nodes,

Nervous system, and

• Extremities.

The number and percentage of subjects with physical examination results by body system classified as

'Normal', 'Abnormal, NCS' or 'Abnormal, CS' will be summarized (Baseline and scheduled visits only).

Shift from Baseline of the physical examination category will also be summarized by body system.


By-subject listing will be provided for subjects who have at least one abnormal result from any body system

or who missed the assessment due to any reason.

All physical examination results will be listed on the Safety population.

13.6. Respiratory Assessments

13.6.1. Asthma Control Test

Subjects with a medical history of asthma will take an Asthma Control Test (ACT) at Baseline/Day 1, Week

4, Week 8, Week 12, Week 16, Week 20 and Week 24, Early Termination visit, and Week 32/Follow-up.

Subjects with new (de novo) diagnosis of asthma will complete the ACT testing beginning from new (de

novo) diagnosis and at all subsequent scheduled visits.

The ACT is composed of 5 questions. For each question, the subject will choose the best answer out of 5

possible answers. The test provides a numerical score ranging from 5 to 25 to assess asthma control; a

higher score indicates better asthma control while a score of 19 or less indicates the subject's asthma may

not be under control.

ACT total score (absolute values and change from Baseline) will be summarized as a continuous variable

(Baseline and scheduled visits only).

The number and percentage of subjects with an ACT score ≤ 19 will be summarized (scheduled visits only).

The ACT results and the ACT score will be listed on the Safety population.

13.6.2. Respiratory Examination

A respiratory examination consists of medical interview. Questions regarding medical history of asthma,

wheeze, dyspnea, and cough, will be performed for all subjects at Baseline/Day 1, Week 12, Week 24,

Early Termination and Week 32/Follow-up questions are asked regarding:

newly diagnosed (de novo) with Asthma / experience a worsening of Asthma since last visit

newly diagnosed with Wheeze since last visit / experience a worsening of Wheeze since last visit

newly diagnosed with Dyspnea since last visit / experience a worsening of Dyspnea since last visit

newly diagnosed with Cough since last visit / experience a worsening of Cough since last visit

Only subjects reporting a medical history of asthma will require a respiratory examination at all visits.

Subjects with a new (de novo) diagnosis of asthma will require a respiratory examination at all scheduled

visits after the diagnosis is first made.


Newly diagnosed asthma or unexpected worsening of asthma are also reported as AESI. Respiratory

examination questionnaire results will be listed on the Safety population.

13.6.3. Peak Expiratory Flow

Peak expiratory flow (PEF) testing during the clinical study will be performed under the supervision of

qualified study personnel. Peak expiratory flow measurements should consist of 3 good efforts, with the

best result documented. Obtained PEF values will be compared to predicted values based on the subject's

age, sex and height.

PEF testing will be performed for all subjects at Baseline/Day 1, Week 12, Week 24, Early Termination, and

Week32/Follow-up visits. For subjects reporting a medical history of asthma, PEF testing will be performed

at all visits during the clinical study. For subjects diagnosed with new (de novo) asthma, PEF testing will be

performed at all visits, starting with the visit in which the diagnosis was confirmed.

Following PEF parameters will be summarized as a continuous variable (Baseline and scheduled visits

only):

Actual peak expiratory flow rate

Predicted peak expiratory flow rate

• Actual PEF of predicted value (%).

These PEF parameters will be summarized separately for the subset of subjects with and without history

of asthma.

The number and percentage of subjects with PEF < 80% will be summarized by treatment group, visit

(baseline and scheduled visits only), and medical history of asthma (with and without history of asthma).

All PEF results will be listed on the Safety population.

# 14. Changes from Analysis Planned in Protocol

• Summary Statistics will be presented by Treatment Group instead of "by Treatment Group and dosing regimen".

## 15. Programming Considerations

All TFLs and statistical analyses will be generated using SAS® 9.4 or higher (SAS® Institute Inc., Cary, NC, USA) on a SAS Server. Changes to the software version (e.g. upgrades), or use of additional software consistent with the SAP will not be considered a violation of the SAP.

#### 15.1. General Considerations

All TFLs will be produced in accordance to CCI (see Section 16).

- A separate SAS program will be created for each output.
- Each output will be stored in a separate file.
- Output files will be provided in separate Word rtf and as combined PDF format including all outputs in one PDF file.
- Numbering of TFLs will follow International Conference on Harmonization (ICH) E3 Guidance.

#### 15.2. Table, Figure, and Listing Format

#### 15.2.1. General

- All TFLs will be produced in landscape format, unless otherwise specified.
- All TFLs will be produced on paper size A4 using the Courier New font, size 8.
- The data displays for all TFLs will have a 1 inch binding margin on top and bottom of a landscape oriented page and a minimum 1.25 inch margin on the left side and a minimum of 0.75 inch right side.
- Headers and footers for figures will be in Courier New font, size 8.
- Legends will be used for all figures with more than 1 variable, group, or item displayed.
- TFLs will be in black and white (no colour), unless otherwise specified.
- Specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text, will not be used in the TFLs, unless otherwise specified. On some occasions, superscripts 1, 2, or 3 may be used (see below).
- Only standard keyboard characters will be used in the TFLs. Special characters, such as non-printable control characters, printer-specific, or font-specific characters, will not be used.


Hexadecimal-derived characters will be used, where possible, if they are appropriate to help display math symbols (e.g.,  $\mu$ ). Certain subscripts and superscripts (e.g., cm2, Cmax) will be employed on

a case-by-case basis.

Mixed case will be used for all titles, footnotes, column headers, and programmer-supplied formats,

as appropriate.

15.2.2. Headers

• All output should have the following header at the top left of each page:

Galderma Protocol RD.06.SPR.203890

Dry-run/Draft/Final

 All output should have Page n of N at the top corner of each page. TFLs are internally paginated in relation to the total length (i.e., the page number should appear sequentially as page n of N, where

N is the total number of pages in the table).

• The date output was generated should appear along with the program name as a footer on each

page.

15.2.3. Display Titles

Each TFL are identified by the designation and a numeral. (i.e., Table 14.1.1.1). ICH E3 numbering

is used. A decimal system (x.y and x.y.z) are used to identify TFLs with related contents. The title

is centered. The analysis population are identified on the line immediately following the title. The

title and table designation are single spaced. A solid line spanning the margins will separate the

display titles from the table.

Column headers. There will be 1 blank line between the last title and the solid line.

Table 14.1.1.1

Screened Population

Subject

15.2.4. Column Headers

Column headings are displayed immediately below the solid line described above in Initial upper-

case characters.

In the case of efficacy tables, the variable (or characteristic) column will be on the far left followed

by the treatment group column.

For numeric variables, include "unit" in column or row heading when appropriate.

Disposition

• Analysis population sizes will be presented for dose group in the column heading as "N=XX" (or in the row headings, if applicable). This is distinct from the 'n' used for the descriptive statistics

representing the number of subjects in the analysis population.

15.2.5. Body of the Data Display

15.2.5.1. General Conventions

Data in columns of a table or listing are formatted as follows:

Alphanumeric values will be left-justified;

• Whole numbers (e.g., counts) will be right-justified; and

Numbers containing fractional portions will be decimal aligned. The "%" is not presented for example

"5 (0.6)"

15.2.5.2. Table Conventions

• Units will be included where available

• If the categories of a parameter are ordered, then all categories between the maximum and minimum

category are presented in the table, even if n=0 for all treatment groups in a given category that is between the minimum and maximum level for that parameter. For example, the frequency distribution

for symptom severity would appear as:

| Severity | N |
|----------|---|
| Rating | |
| severe | 0 |
| moderate | 8 |
| mild | 3 |

Where percentages are presented in these tables, zero percentages will not be presented and so counts of 0 will be presented as 0 and not as 0 (0).

• If the categories are not ordered (e.g., Medical History, Reasons for Discontinuation from the Study,

etc.), then only those categories for which there is at least 1 subject represented are included.

An Unknown or Missing category will be added to each parameter for which information is not

available for 1 or more subjects

 Unless otherwise specified, the estimated mean, median, Q1 and Q3 for a set of values are printed out to 1 more significant digit than the original values, and standard deviations are printed out to 2

more significant digits than the original values. The minimum and maximum should report the same


significant digits as the original values. Missing descriptive statistics or p-values which cannot be

estimated are reported as "-".

• Percentage values will be printed to one decimal place without the "%", with the "." in alignment, one

space after the count (e.g., 7 (12.8), 13 (5.4)). Unless otherwise noted, for all percentages, the

number of subjects in the analysis set for the treatment group who have an observation will be the

denominator. Percentages after zero counts will not be displayed and percentages equating to 100%

will be presented as 100, without decimal places.

• Tabular display of data for medical history, prior/concomitant medications, and all tabular displays of

adverse event data are presented by the body system, treatment class, or SOC. The body system,

drug class and SOC are displayed in alphabetically order. Within body system, drug class and SOC,

preferred term will be display in descending frequency. If incidence for more than 1 preferred term is

identical, they should then be sorted alphabetically.

P-values will be output in the format: '0.xxxx', where xxx is the value rounded to 4 decimal places.

Every p-value less than 0.0001 will be presented as "<0.0001". If the p-value is returned as >0.9999,

then present as ">0.9999".

• The percentage of subjects is normally calculated as a proportion of the number of subjects assessed

in the relevant treatment group (or overall) for the analysis population presented. However, careful

consideration is required in many instances due to the complicated nature of selecting the

denominator, usually the appropriate number of subjects exposed. These details are described in

footnotes or programming notes.

For categorical summaries (number and percentage of subjects) where a subject can be included in

more than one category, it is described in a footnote or programming note as needed if the subject

are included in the summary statistics for all relevant categories or just 1 category and the criteria for

selecting the criteria.

Where a category with a subheading (such as system organ class) has to be split over more than

one page, output the subheading followed by "(cont.)" at the top of each subsequent page. The

overall summary statistics for the subheading should only be output on the first relevant page.

**15.2.5.3.** Listing Conventions

• Listings will be sorted for presentation in order of subject number, visit/collection day, and

visit/collection time.


• Missing data will be represented on subject listings as either a hyphen ('-') with a corresponding

footnote ('- = unknown or not evaluated'), or as 'N/A', with the footnote 'N/A = not applicable',

whichever is appropriate.

Dates will be printed in SAS DATE9.format ('DD\_MMM\_YYYY': 01JUL2000). Missing portions of

dates will be represented on subject listings as dashes (--JUL2000). Dates that are missing because

they are not applicable for the subject will be output as 'N/A', unless otherwise specified.

• All observed time values will be presented using a 24-hour clock HH:MM or HH:MM:SS format (e.g.,

11:26:45, or 11:26). Time will only be reported if it was measured as part of the study.

• Units will be included where available.

**15.2.5.4.** Figure Conventions

• Unless otherwise specified, for all figures, study visits will be displayed on the X-axis and endpoint

(e.g., treatment mean change from Baseline) values will be displayed on the Y-axis.

15.2.6. Footnotes

• A solid line spanning the margins will separate the body of the data display from the footnotes.

• All footnotes will be left justified with single-line spacing immediately below the solid line underneath

the data display.

• Footnotes will always begin with 'Notes:' if an informational footnote, or 1, 2, 3, etc. if a reference

footnote. Each new footnote will start on a new line, where possible.

Subject specific footnotes are avoided, where possible.

Footnotes will be used sparingly and add value to the TFL. If more than 10 lines of footnotes are

planned, then a cover page is strongly recommended to be used to display footnotes, and only those

essential to comprehension of the data will be repeated on each page.

• The last line of the footnote section will be a standard source line that indicates the name of the

program used to produce the data display, date the program was run, the date of extraction indicated

with "Data Cut-off: DDMMMYYYY" and the listing source (i.e., 'Program: t-14-01-03-02-01.sas,

Run date: 16MAR2021 12:57', date cut-off: DDMMMYYYY, Listing Source(s): 16.x.y.z).

Sources and/or cross-references in footnotes will use the keyword prefix (in singular form) for each

reference and will be separated by a comma when multiple cross-references are displayed.

Statistical Analysis Plan for Interventional Studies

## **Example**

Listing source: 16.2.1.1

## 16. Quality Control

SAS programs are developed to produce output such as analysis data sets, summary tables, data listings, figures or statistical analyses. An overview of the development of programs is detailed in CCI Developing Statistical Programs Standard Operation Procedure (SOP) (3907).

SOPs Developing Statistical Programs (3907) and Conducting the Transfer of Biostatistical Deliverables (SDTM, ADaM, TFL) (3908) describes the quality control procedures that are performed for all SAS programs and output. Quality control is defined here as the operational techniques and activities undertaken to verify that the SAS programs produce the output by checking for their logic, efficiency and commenting and by review of the produced output. A detailed description of project specific QC procedure can be found in the document "SAS Programming and Validation Plan".

## 17. Index of Tables

This section contains lists of the tables tentatively planned for this study. Changes in the number or content of planned listings are not considered deviations from this SAP.

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| 14. | | TABLES AND FIGURES | |
| 14.1 | | Demographic Data | |
| 14.1.1 | | Subject Disposition | |
| | 14.1.1.1 | Subject Accounting by Overall, Country and | ITT Population |
| | | Site | |
| | 14.1.1.2 | Subject Accounting by Visit | ITT Population |
| | 14.1.1.3 | Summary of Subject Disposition | ITT Population |
| | 14.1.1.4 | Summary of Subject Disposition by Site | ITT Population |
| | 14.1.1.5 | Summary of Analysis Populations | ITT Population |
| 14.1.2 | | Protocol Deviations | |
| | 14.1.2.1 | Summary of Major Protocol Deviations | ITT Population |
| | 14.1.2.2 | Summary of Major Protocol Deviations by | ITT Population |
| | | Site | |
| 14.1.3 | | Demographic and Baseline Characteristics | |
| 14.1.3.1 | | Subject Demographic and Baseline | |
| | | Characteristics | |
| | 14.1.3.1.1 | Subject Demographic and Baseline | ITT Population |
| | | Characteristics | |
| | 14.1.3.1.2 | Subject Demographic and Baseline | Safety Population |
| | | Characteristics | |
| | 14.1.3.1.3 | Subject Demographic and Baseline | Per-Protocol |
| | | Characteristics | Population |
| | 14.1.3.1.4 | Subject Demographic and Baseline | POE Analysis |
| | | Characteristics | Population |
| 14.1.3.2 | | Baseline Disease Characteristics | |
| | 14.1.3.2.1 | Summary of Baseline Disease | ITT Population |
| | | Characteristics | |
| | 14.1.3.2.2 | Summary of Baseline Disease | Safety Population |
| | | Characteristics | |

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| | 14.1.3.2.3 | Summary of Baseline Disease | Per-Protocol |
| | | Characteristics | Population |
| | 14.1.3.2.4 | Summary of Baseline Disease | POE Analysis |
| | | Characteristics | Population |
| | 14.1.3.2.5 | Summary of Proportion of Subjects with | ITT Population |
| | | Differences between Randomization | |
| | | Stratification and Actual Stratification | |
| 14.1.3.3 | | Medical History | |
| | 14.1.3.3.1 | Summary of Previous and Ongoing Medical | ITT Population |
| | | History | |
| | 14.1.3.3.2 | Summary of Prior Medical and Surgical | ITT Population |
| | | Procedures | |
| | 14.1.3.3.3 | Summary of Concomitant Medical and | ITT Population |
| | | Surgical Procedures during Treatment | |
| | | Period | |
| | 14.1.3.3.4 | Summary of Concomitant Medical and | ITT Population |
| | | Surgical Procedures during Follow-up | |
| | | Period | |
| 14.1.4 | | Medications | |
| | 14.1.4.1 | Summary of Prior Medications by ATC level | ITT Population |
| | | and Preferred Term | |
| | 14.1.4.2 | Summary of Concomitant Medications | ITT Population |
| | | during Treatment Period by ATC level and | |
| | | Preferred Term | |
| | 14.1.4.3 | Summary of Concomitant Medications | ITT Population |
| | | during Follow-up Period by ATC level and | |
| | | Preferred Term | |
| | 14.1.4.4 | Summary of Prohibited Medications during | ITT Population |
| | | Treatment Period by ATC level and | |
| | | Preferred Term | |
| | 14.1.4.5 | Summary of Prohibited Medications during | ITT Population |
| | | Follow-up Period by ATC level and Preferred | |
| | | Term | |
| 14.1.5 | | Treatment Compliance | |

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| | 14.1.5.1 | Summary of Exposure to Study Drug | Safety Population |
| 14.2 | | Efficacy Data | |
| 14.2.1 | | Primary Efficacy Parameters | |
| | 14.2.1.1.1 | Time to Relapse | ITT Population |
| | 14.2.1.1.3 | | Per-Protocol |
| | | Sensitivity Analysis of Time to Relapse | Population |
| | 14.2.1.1.5 | Sensitivity Analysis of Time to Relapse - | ITT Population |
| | | using Actual Stratifications | |
| | 14.2.1.1.7 | Sensitivity Analysis of Time to Relapse - | ITT Population |
| | | Removing COVID-19 affected Visits | |
| 14.2.2 | | Secondary Efficacy Parameters | |
| 14.2.2.1 | | Secondary Efficacy Parameter: IGA | |
| | 14.2.2.1.1 | Summary of IGA - OC | ITT Population |
| | 14.2.2.1.2 | | Per-Protocol |
| | | Summary of IGA - OC | Population |
| | 14.2.2.1.3 | Summary of Proportion of Subjects with | ITT Population |
| | | maintaining IGA Success - OC | |
| | 14.2.2.1.4 | Analysis of Proportion of Subjects with | ITT Population |
| | | maintaining IGA Success – OC | |
| | 14.2.2.1.5 | Analysis of Proportion of Subjects with | Per-Protocol |
| | | maintaining IGA Success – OC | Population |
| | 14.2.2.1.6 | Analysis of Proportion of Subjects with | ITT Population |
| | | maintaining IGA Success - Missing as non- | |
| | | responder | |
| | 14.2.2.1.8 | Summary of Proportion of Subjects with | ITT Population |
| | | increase in IGA >= 2 points from baseline - | |
| | | oc | |
| | 14.2.2.1.9 | Analysis of Proportion of Subjects with | ITT Population |
| | | increase in IGA >= 2 points from baseline - | |
| | | ос | |
| | 14.2.2.1.10 | Analysis of Proportion of Subjects with | Per-Protocol |
| | | increase in IGA >= 2 points from baseline - | Population |
| | | ос | |

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| | 14.2.2.1.11 | Analysis of Proportion of Subjects with | ITT Population |
| | | increase in IGA >= 2 points from baseline - | |
| | | Missing as non-responder | |
| 14.2.2.2 | | Secondary Efficacy Parameter: Peak | |
| | | Pruritus Numeric Rating Scale | |
| | 14.2.2.2.1 | Summary of Weekly PP NRS – OC | ITT Population |
| | 14.2.2.2.2 | | Per-Protocol |
| | | Summary of Weekly PP NRS - OC | Population |
| | 14.2.2.2.3 | Summary of Proportion of Subjects with | ITT Population |
| | | Weekly PP NRS increase >= 4 | |
| | 14.2.2.2.4 | Analysis of Proportion of subjects with | ITT Population |
| | | increase in PP NRS score >= 4 points from | |
| | | baseline - OC | |
| | 14.2.2.2.5 | Analysis of Proportion of subjects with | Per-Protocol |
| | | increase in PP NRS score >= 4 points from | Population |
| | | baseline – OC | |
| | 14.2.2.2.6 | Analysis of Proportion of subjects with | ITT Population |
| | | increase in PP NRS score >= 4 points from | |
| | | baseline – Missing as non-responder | |
| | 14.2.2.2.7 | Analysis of Change from Baseline in Weekly | ITT Population |
| | | PP NRS at Weeks 4, 8, 12, 16, 20 and 24 - | |
| | | OC - ANCOVA | |
| | 14.2.2.2.8 | Analysis of Change from Baseline in Weekly | Per-Protocol |
| | | PP NRS at Weeks 4, 8, 12, 16, 20 and 24 - | Population |
| | | OC - ANCOVA | |
| | 14.2.2.2.9 | Analysis of Change from Baseline for | ITT Population |
| | | Weekly PP NRS at Weeks 4, 8, 12, 16, 20 | |
| | | and 24 – MMRM Analysis | |
| 14.2.2.3 | | Secondary Efficacy Parameter: Sleep | |
| | | Disturbance Numeric Rating Scale | |
| | 14.2.2.3.1 | Summary of Weekly SD NRS - OC | ITT Population |
| | 14.2.2.3.2 | | Per-Protocol |
| | | Summary of Weekly SD NRS - OC | Population |
| | 14.2.2.3.3 | Analysis of Change from Baseline in Weekly | ITT Population |
| | | SD NRS - ANCOVA | |

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| | 14.2.2.3.4 | Analysis of Change from Baseline in Weekly | Per-Protocol |
| | | SD NRS - ANCOVA | Population |
| | 14.2.2.3.5 | Analysis of Change from Baseline for | ITT Population |
| | | Weekly SD NRS – MMRM Analysis | |
| 14.2.2.4 | | Secondary Efficacy Parameter: | |
| | | Dermatology Life Quality Index | |
| | 14.2.2.4.1 | Summary of DLQI – OC | ITT Population |
| | 14.2.2.4.2 | Analysis of Change from Baseline in DLQI - | ITT Population |
| | | OC – ANCOVA | |
| 14.2.3 | | Pharmacokinetics | |
| | 14.2.3.1 | Summary of Nemolizumab Serum | POE Population |
| | | Concentrations | |
| 14.2.4 | | Immunogenicity | |
| | 14.2.4.1 | Summary of Immunogenicity - Anti-drug | POE Population |
| | | Antibody (ADA) and Neutralizing Antibody | |
| 14.3 | | Safety Data Summary Tables | |
| 14.3.1 | | Adverse Events | |
| | 14.3.1.1.1 | Overall Summary of Treatment Emergent | Safety Population |
| | | Adverse Events (TEAEs) during Treatment | |
| | | Period, All Causalities | |
| | 14.3.1.1.2 | Overall Summary of Treatment Emergent | Safety Population |
| | | Adverse Events (TEAEs) during Follow-up | |
| | | Period, All Causalities | |
| | 14.3.1.1.3 | Overall Summary of Treatment Emergent | Safety Population |
| | | Adverse Events (TEAEs) during Overall | |
| | | Study Period, All Causalities | |
| | 14.3.1.1.4 | Overall Summary of Treatment Emergent | Safety Population |
| | | Adverse Events (TEAEs) during Treatment | |
| | | Period, Study Drug Related | |
| | 14.3.1.1.5 | Overall Summary of Treatment Emergent | Safety Population |
| | | Adverse Events (TEAEs) during Follow-up | |
| | | Period, Study Drug Related | |

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| | 14.3.1.1.6 | Overall Summary of Treatment Emergent | Safety Population |
| | | Adverse Events (TEAEs) during Overall | |
| | | Study Period, Study Drug Related | |
| | 14.3.1.1.7 | Overall Summary of Treatment Emergent | Safety Population – |
| | | Adverse Events (TEAEs) during Treatment | Subjects with |
| | | Period, All Causalities | COVID-19 Infection |
| | 14.3.1.1.8 | Overall Summary of Treatment Emergent | Safety Population – |
| | | Adverse Events (TEAEs) during Follow-up | Subjects with |
| | | Period, All Causalities | COVID-19 Infection |
| | 14.3.1.1.9 | Overall Summary of Treatment Emergent | Safety Population – |
| | | Adverse Events (TEAEs) during Treatment | Subjects with |
| | | Period, Study Drug Related | COVID-19 Infection |
| | 14.3.1.1.10 | Overall Summary of Treatment Emergent | Safety Population – |
| | | Adverse Events (TEAEs) during Follow-up | Subjects with |
| | | Period, Study Drug Related | COVID-19 Infection |
| | 14.3.1.2.1 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) during Treatment Period by SOC | |
| | | and PT, All Causalities | |
| | 14.3.1.2.2 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) during Follow-up Period by SOC | |
| | | and PT, All Causalities | |
| | 14.3.1.2.3 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) during Overall Study Period by | |
| | | SOC and PT, All Causalities | |
| | 14.3.1.2.4 | Treatment Emergent Adverse Events | Safety Population – |
| | | (TEAEs) during Treatment Period by SOC | Subjects with |
| | | and PT, All Causalities | COVID-19 Infection |
| | 14.3.1.2.5 | Treatment Emergent Adverse Events | Safety Population – |
| | | (TEAEs) during Follow-up Period by SOC | Subjects with |
| | | and PT, All Causalities | COVID-19 Infection |
| | 14.3.1.3.1 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) during Treatment Period by SOC | |
| | | and PT, Study Drug Related | |

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| | 14.3.1.3.2 | Treatment Emergent Adverse Events (TEAEs) during Follow-up Period by SOC | Safety Population |
| | | and PT, Study Drug Related | |
| | 14.3.1.3.3 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) during Overall Study Period by SOC and PT, Study Drug Related | |
| | 14.3.1.3.4 | Treatment Emergent Adverse Events | Safety Population – |
| | | (TEAEs) during Treatment Period by SOC | Subjects with |
| | | and PT, Study Drug Related | COVID-19 Infection |
| | 14.3.1.3.5 | Treatment Emergent Adverse Events | |
| | | (TEAEs) during Follow-up Period by SOC | Subjects with |
| | | and PT, Study Drug Related | COVID-19 Infection |
| | 14.3.1.4 | Exposure-Adjusted Incidence Rate for | Safety Population |
| | | Treatment Emergent Adverse Events | |
| | | (TEAEs) during Treatment Period by SOC | |
| | | and PT, All Causalities | |
| | 14.3.1.5 | Exposure-Adjusted Incidence Rate of | Safety Population |
| | | Treatment Emergent Adverse Events | |
| | | (TEAEs) during Treatment Period by SOC | |
| | | and PT, Study Drug Related | |
| | 14.3.1.6.1 | Serious Treatment Emergent Adverse | Safety Population |
| | | Events (TEAEs) during Treatment Period by | |
| | | SOC and PT, All Causalities | |
| | 14.3.1.6.2 | Serious Treatment Emergent Adverse | |
| | | Events (TEAEs) during Follow-up Period by | |
| | | SOC and PT, All Causalities | |
| | 14.3.1.6.3 | Serious Treatment Emergent Adverse | Safety Population – |
| | | Events (TEAEs) during Treatment Period by | Subjects with |
| | | SOC and PT, All Causalities | COVID-19 Infection |
| | 14.3.1.6.4 | Serious Treatment Emergent Adverse | Safety Population – |
| | | Events (TEAEs) during Follow-up Period by | Subjects with |
| | | SOC and PT, All Causalities | COVID-19 Infection |
| | 14.3.1.7.1 | Serious Treatment Emergent Adverse | Safety Population |
| | | Events (TEAEs) during Treatment Period by | |
| | | SOC and PT, Study Drug Related | |
| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| | 14.3.1.7.2 | Serious Treatment Emergent Adverse | Safety Population |
| | | Events (TEAEs) during Follow-up Period by | |
| | | SOC and PT, Study Drug Related | |
| | 14.3.1.7.3 | Serious Treatment Emergent Adverse | Safety Population – |
| | | Events (TEAEs) during Treatment Period by | Subjects with |
| | | SOC and PT, Study Drug Related | COVID-19 Infection |
| | 14.3.1.7.4 | Serious Treatment Emergent Adverse | Safety Population – |
| | | Events (TEAEs) during Follow-up Period by | Subjects with |
| | | SOC and PT, Study Drug Related | COVID-19 Infection |
| | 14.3.1.8 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) during Treatment Period by SOC, | |
| | | PT and Maximum Severity, All Causalities | |
| | 14.3.1.8.2 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) during Follow-up Period by SOC, | |
| | | PT and Maximum Severity, All Causalities | |
| | 14.3.1.9.1 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) during Treatment Period by SOC, | |
| | | PT and Maximum Severity, Study Drug | |
| | | Related | |
| | 14.3.1.9.2 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) during Follow-up Period by SOC, | |
| | | PT and Maximum Severity, Study Drug | |
| | | Related | |
| | 14.3.1.10.1 | Severe Treatment Emergent Adverse | Safety Population |
| | | Events (TEAEs) during Treatment Period by | |
| | | SOC and PT, All Causalities | |
| | 14.3.1.10.2 | Severe Treatment Emergent Adverse | Safety Population |
| | | Events (TEAEs) during Follow-up Period by | |
| | | SOC and PT, All Causalities | |
| | 14.3.1.11.1 | Severe Treatment Emergent Adverse | Safety Population |
| | | Events (TEAEs) during Treatment Period by | |
| | | SOC and PT, Study Drug Related | |
| | 14.3.1.11.2 | Severe Treatment Emergent Adverse | Safety Population |
| | | Events (TEAEs) during Follow-up Period by | |
| | | SOC and PT, Study Drug Related | |
| | | Joo and Fr, Study Drug Related | |

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| | 14.3.1.12.1 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) Leading to Permanent | |
| | | Discontinuation of Study Drug during | |
| | | Treatment Period by SOC and PT, All | |
| | | Causalities | |
| | 14.3.1.13.1 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) Leading to Permanent | |
| | | Discontinuation of Study Drug during | |
| | | Treatment Period by SOC and PT, Study | |
| | | Drug Related | |
| | 14.3.1.14.1 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) Leading to Study Discontinuation | |
| | | during Treatment Period by SOC and PT, All | |
| | | Causalities | |
| | 14.3.1.14.2 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) Leading to Study Discontinuation | |
| | | during Follow-up Period by SOC and PT, All | |
| | | Causalities | |
| | 14.3.1.15.1 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) Leading to Study Discontinuation | |
| | | during Treatment Period by SOC and PT, | |
| | | Study Drug Related | |
| | 14.3.1.15.2 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) Leading to Study Discontinuation | |
| | | during Follow-up Period by SOC and PT, | |
| | | Study Drug Related | |
| | 14.3.1.16.1 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) of Special Interest during | |
| | | Treatment Period by Category, SOC and PT, | |
| | | All Causalities | |
| | 14.3.1.16.2 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) of Special Interest during Follow-up | |
| | | Period by Category, SOC and PT, All | |
| | | Causalities | |
| | 1 | I | ı |

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| | 14.3.1.16.3 | Treatment Emergent Adverse Events | Safety Population – |
| | | (TEAEs) of Special Interest during | Subjects with |
| | | Treatment Period by Category, SOC and PT | COVID-19 Infection |
| | 14.3.1.16.4 | Treatment Emergent Adverse Events | Safety Population – |
| | | (TEAEs) of Special Interest during Follow-up | Subjects with |
| | | Period by Category, SOC and PT | COVID-19 Infection |
| | 14.3.1.17.1 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) of Special Interest during | |
| | | Treatment Period by Category, SOC and PT, | |
| | | Study Drug Related | |
| | 14.3.1.17.2 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) of Special Interest during Follow-up | |
| | | Period by Category, SOC and PT, Study | |
| | | Drug Related | |
| | 14.3.1.17.3 | Treatment Emergent Adverse Events | Safety Population – |
| | | (TEAEs) of Special Interest during | Subjects with |
| | | Treatment Period by Category, SOC and PT, | COVID-19 Infection |
| | | Study Drug Related | |
| | 14.3.1.17.4 | Treatment Emergent Adverse Events | Safety Population - |
| | | (TEAEs) of Special Interest during Follow-up | Subjects with |
| | | Period by Category, SOC and PT, Study | COVID-19 Infection |
| | | Drug Related | |
| | 14.3.1.18.1 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) Occurred in PT >= 5% of Subjects | |
| | | during Treatment Period by SOC and PT, All | |
| | | Causalities | |
| | 14.3.1.18.2 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) Occurred in PT >= 5% of Subjects | |
| | | during Follow-up Period by SOC and PT, All | |
| | | Causalities | |
| | 14.3.1.19.1 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) Occurred in PT >= 5% of Subjects | |
| | | during Treatment Period by SOC and PT, | |
| | | Study Drug Related | |

| Table Number | Name | Analysis Set |
|---|---|---|
| 14.3.1.19.2 | Treatment Emergent Adverse Events | Safety Population |
| | (TEAEs) Occurred in PT >= 5% of Subjects | |
| | during Follow-up Period by SOC and PT, | |
| | Study Drug Related | |
| 14.3.1.20.1 | Adjudicated Treatment Emergent Adverse | Safety Population |
| | Events (TEAEs) during Treatment Period by | |
| | SOC and PT, All Causalities | |
| 14.3.1.20.2 | Adjudicated Treatment Emergent Adverse | Safety Population |
| | Events (TEAEs) during Follow-up Period by | |
| | SOC and PT, All Causalities | |
| 14.3.1.21.1 | Adjudicated Treatment Emergent Adverse | Safety Population |
| | Events (TEAEs) during Treatment Period by | |
| | SOC and PT, Study Drug Related | |
| 14.3.1.21.2 | Adjudicated Treatment Emergent Adverse | Safety Population |
| | Events (TEAEs) during Follow-up Period by | |
| | SOC and PT, Study Drug Related | |
| 14.3.1.22.1 | Treatment Emergent Adverse Events | Safety Population |
| | (TEAEs) of Asthma and AESI reported by | |
| | Investigator with Adjudication Outcome | |
| | during Treatment Period by IAC, All | |
| | Causalities | |
| 14.3.1.22.2 | Treatment Emergent Adverse Events | Safety Population |
| | (TEAEs) of Asthma and AESI reported by | |
| | Investigator with Adjudication Outcome | |
| | during Follow-up Period by IAC, All | |
| | Caualities | |
| 14.3.1.23.1 | Treatment Emergent Adverse Events | Safety Population |
| | (TEAEs) of Asthma and AESI reported by | |
| | Investigator with Adjudication Outcome | |
| | during Treatment Period by IAC, Study Drug | |
| | Related | |
| | 14.3.1.20.1<br>14.3.1.20.2<br>14.3.1.21.1<br>14.3.1.21.2<br>14.3.1.22.1 | Treatment Emergent Adverse Events (TEAEs) Occurred in PT >= 5% of Subjects during Follow-up Period by SOC and PT, Study Drug Related 14.3.1.20.1 Adjudicated Treatment Emergent Adverse Events (TEAEs) during Treatment Period by SOC and PT, All Causalities 14.3.1.20.2 Adjudicated Treatment Emergent Adverse Events (TEAEs) during Follow-up Period by SOC and PT, All Causalities 14.3.1.21.1 Adjudicated Treatment Emergent Adverse Events (TEAEs) during Treatment Period by SOC and PT, Study Drug Related 14.3.1.21.2 Adjudicated Treatment Emergent Adverse Events (TEAEs) during Follow-up Period by SOC and PT, Study Drug Related 14.3.1.22.1 Treatment Emergent Adverse Events (TEAEs) of Asthma and AESI reported by Investigator with Adjudication Outcome during Treatment Emergent Adverse Events (TEAEs) of Asthma and AESI reported by Investigator with Adjudication Outcome during Follow-up Period by IAC, All Causalities 14.3.1.23.1 Treatment Emergent Adverse Events (TEAEs) of Asthma and AESI reported by Investigator with Adjudication Outcome during Follow-up Period by IAC, All Caualities 14.3.1.23.1 Treatment Emergent Adverse Events (TEAEs) of Asthma and AESI reported by Investigator with Adjudication Outcome during Follow-up Period by IAC, All Caualities |

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| | 14.3.1.23.2 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) of Asthma and AESI reported by | |
| | | Investigator with Adjudication Outcome | |
| | | during Treatment Period by IAC, Study Drug | |
| | | Related | |
| | 14.3.1.24.1 | Confirmed Adjudicated Treatment Emergent | Safety Population |
| | | Adverse Events (TEAEs) during Treatment | |
| | | Period by SOC, PT and Maximum Severity, | |
| | | All Causalities | |
| | 14.3.1.24.2 | Confirmed Adjudicated Treatment Emergent | Safety Population |
| | | Adverse Events (TEAEs) during Follow-up | |
| | | Period by SOC, PT and Maximum Severity, | |
| | | All Causalities | |
| | 14.3.1.25.1 | Confirmed Adjudicated Treatment Emergent | Safety Population |
| | | Adverse Events (TEAEs) during Treatment | |
| | | Period by SOC, PT and Maximum Severity, | |
| | | Study Drug Related | |
| | 14.3.1.25.2 | Confirmed Adjudicated Treatment Emergent | Safety Population |
| | | Adverse Events (TEAEs) during Follow-up | |
| | | Period by SOC, PT and Maximum Severity, | |
| | | Study Drug Related | |
| | 14.3.1.26.1 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) of Special Interest during | |
| | | Treatment Period by Category, SOC, PT and | |
| | | Maximum Severity, All Causalities | |
| | 14.3.1.26.2 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) of Special Interest during Follow-up | |
| | | Period by Category, SOC, PT and Maximum | |
| | | Severity, All Causalities | |
| | 14.3.1.27.1 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) of Special Interest during | |
| | | Treatment Period by Category, SOC, PT and | |
| | | Maximum Severity, Study Drug Related | |
| | L | | |

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| | 14.3.1.27.2 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAEs) of Special Interest during Follow-up | |
| | | Period by Category, SOC, PT and Maximum | |
| | | Severity, Study Drug Related | |
| 14.3.2 | | Listings of Deaths, Other Serious and | |
| | | Significant Adverse Events | |
| | 14.3.2.1 | Listing of Serious Treatment Emergent | Safety Population |
| | | Adverse Events (TEAEs) | |
| | 14.3.2.2 | Listing of Severe Treatment Emergent | Safety Population |
| | | Adverse Events (TEAEs) | |
| | 14.3.2.3 | Listing of Treatment Emergent Adverse | Safety Population |
| | | Events (TEAEs) Leading to Permanent | |
| | | Discontinuation of Study Drug | |
| | 14.3.2.4 | Listing of Treatment Emergent Adverse | Safety Population |
| | | Events (TEAEs) of Special Interest | |
| | 14.3.2.5 | Listing of Treatment Emergent Adverse | Safety Population |
| | | Events (TEAEs) Leading to Death | |
| 14.3.3 | | Narratives of Deaths, Other Serious and | |
| | | Certain Other Significant Adverse Events | |
| 14.3.4 | | Laboratory Value | |
| 14.3.4.1 | | Clinical Laboratory Data | |
| 14.3.4.1.1 | | Hematology Data | |
| | 14.3.4.1.1.1 | Summary of Laboratory Data for | Safety Population |
| | | Hematology | |
| | 14.3.4.1.1.2 | Shift from Baseline for Hematology by | Safety Population |
| | | Reference Ranges | |
| | 14.3.4.1.1.3 | Summary of Potentially Clinically Significant | Safety Population |
| | | Hematology | |
| | 14.3.4.1.1.4 | Listing of Subjects with Abnormal | Safety Population |
| | | Hematology Results | |
| | 14.3.4.1.1.5 | Listing of Subjects with Potentially Clinically | Safety Population |
| | | Significant Hematology Results | |
| 14.3.4.1.2 | | Blood Chemistry Data | |
| | 14.3.4.1.2.1 | Summary of Laboratory Data for Clinical | Safety Population |
| | | Chemistry | |
| | | ı | |

| Safety Population |
|---|
| Safety Population Safety Population Safety Population Safety Population Safety Population |
| Safety Population Safety Population Safety Population Safety Population Safety Population |
| Safety Population Safety Population Safety Population Safety Population |
| Safety Population Safety Population Safety Population Safety Population |
| Safety Population Safety Population Safety Population |
| Safety Population Safety Population Safety Population |
| Safety Population Safety Population |
| Safety Population Safety Population |
| Safety Population Safety Population |
| Safety Population |
| Safety Population |
| Safety Population |
| Salety Fubulation |
| Safety Population |
| Safety Population |
| Safety Population |
| Safety Population |
| Safety Population |
| Safety Population |
| Safety Population |
| Safety Population |
| Safety Population |

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| | 14.3.4.4.6 | Summary of Respiratory Assessments - | Safety Population |
| | | Peak Expiratory Flow (PEF) for Subjects | |
| | | without Asthma History | |
| | 14.3.4.4.7 | Summary of Peak Expiratory Flow (PEF) < | Safety Population |
| | | 80% of Predicted Value | |
| | 14.3.4.4.8 | Summary of Peak Expiratory Flow (PEF) < | Safety Population |
| | | 80% of Predicted Value for Subjects with | |
| | | Asthma History | |
| | 14.3.4.4.9 | Summary of Peak Expiratory Flow (PEF) < | Safety Population |
| | | 80% of Predicted Value for Subjects without | |
| | | Asthma History | |
| | 14.3.4.4.10 | Summary of Asthma Control Test (ACT) | Safety Population |
| | 14.3.4.4.11 | Summary of Respiratory Examination | Safety Population |

## 18. Index of Figures

This section contains lists of the figures tentatively planned for this study. Changes in the number or content of planned listings are not considered deviations from this SAP.

| Figure | Name | Analysis Set |
|---|---|---|
| Number | | (Examples) |
| 14.1.1.5 | Time (days) to Permanent Discontinuation of Study Drug by Reason | ITT Population |
| | for Discontinuation | |
| 14.2.1.1.2 | KM Plot - Time to Relapse | ITT Population |
| 14.2.1.1.4 | KM Plot - Time to Relapse | Per-Protocol |
| | | Population |
| 14.2.1.1.6 | KM Plot - Time to Relapse – using Actual Stratification | ITT Population |
| 14.2.1.1.8 | KM Plot - Time to Relapse – Removing COVID-19 affected visits | ITT Population |
| 14.2.2.1.7 | Line Plot of Proportion of Subjects with maintaining IGA Success – | ITT Population |
| | Missing as Non-Responder | |
| 14.2.2.1.12 | Line Plot of Proportion of Subjects with increase in IGA >= 2 points | ITT Population |
| | from baseline – Missing as Non-Responder | |
| 14.2.2.2.7 | Line Plot of Proportion of Subjects with increase in Weekly Average | ITT Population |
| | PP NRS >= 4 - Missing as Non-Responder | |
| 14.2.3.2 | Mean Nemolizumab Time-Concentration Profiles | POE Analysis |
| | | Population |
| 14.2.3.3 | Individual Time-Concentration Profiles | POE Analysis |
| | | Population |
| 14.3.4.1.1.6 | Distribution of Hematology Laboratory Parameters by Visit with | Safety |
| | Maximum Post-Baseline Values | Population |
| 14.3.4.1.2.6 | Distribution of Chemistry Laboratory Parameters by Visit with | Safety |
| | Maximum Post-Baseline Values | Population |
| 14.3.4.2.4 | Distribution of Vital Signs by Visit with Maximum Post-baseline | Safety |
| | Values | Population |

# 19. Index of Listings

This section contains lists of the listings tentatively planned for this study. Changes in the number or content of planned listings are not considered deviations from this SAP.

| | Listing | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| 16.2 | | Subject Data Listings | |
| 16.2.1 | | Discontinued Subjects | |
| | 16.2.1.1 | Randomization | ITT Population |
| | 16.2.1.2 | Study Completion Status | ITT Population |
| | 16.2.1.3 | Study Drug Completion Status | ITT Population |
| | 16.2.1.4 | Visit Dates | ITT Population |
| | 16.2.1.5 | Missing Assessment due to COVID-19 | ITT Population |
| 16.2.2 | | Protocol Deviations | |
| | 16.2.2.1 | Protocol Deviations | ITT Population |
| 16.2.3 | | Subjects Excluded from Analysis | |
| | | Populations | |
| | 16.2.3.1 | Subjects in Analysis Populations | ITT Population |
| | 16.2.3.2 | Inclusion and Exclusion Criteria Not Met | All Subjects |
| 16.2.4 | | Demographic Data | |
| | 16.2.4.1 | Demographics and Baseline Characteristics | ITT Population |
| | 16.2.4.2 | Baseline Disease Characteristics | ITT Population |
| | 16.2.4.3 | Medical History | ITT Population |
| | 16.2.4.4 | Medical and Surgical Procedures | ITT Population |
| | 16.2.4.5 | Prior and Concomitant Medications | ITT Population |
| | 16.2.4.6 | Prohibited Medications | ITT Population |
| | 16.2.4.7 | Background Therapy Medications | ITT Population |
| | 16.2.4.8 | Subjects with Difference between | ITT Population |
| | | Randomization Stratification and Actual | |
| | | Stratification | |
| 16.2.5 | | Compliance and Exposure Information | |
| | 16.2.5.1 | Study Drug Dispensation | Safety Population |
| | 16.2.5.2 | Study Drug Administration | Safety Population |
| | 16.2.5.3 | Study Drug Compliance | Safety Population |
| 16.2.6 | | Individual Efficacy Response Data | |

| | Listing | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| | 16.2.6.1 | Time to Relapse | ITT Population |
| | 16.2.6.2 | Investigator's Global Assessment (IGA) | ITT Population |
| | 16.2.6.3 | Pruritus Numeric Rating Scale | ITT Population |
| | 16.2.6.4 | Sleep Disturbance NRS | ITT Population |
| | 16.2.6.5 | Dermatology Life Quality Index (DLQI) | ITT Population |
| | 16.2.6.6 | Nemolizumab Serum Concentrations | POE Analysis |
| | | | Population |
| | 16.2.6.7 | Immunogenicity - Anti-drug Antibody (ADA) | POE Analysis |
| | | and Neutralizing Antibodies | Population |
| 16.2.7 | | Adverse Event Listings | |
| | 16.2.7.1 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAE) | |
| | 16.2.7.2 | Pre-Treatment Adverse Events | Safety Population |
| | 16.2.7.3 | Treatment Emergent Adverse Events | Safety Population |
| | | (TEAE) Comments | |
| | 16.2.7.4 | Adjudicated Asthma Treatment Emergent | Safety Population |
| | | Adverse Events (TEAE) | |
| | 16.2.7.5 | Adjudicate Asthma Treatment Emergent | Safety Population |
| | | Adverse Events (TEAE) Comments by | |
| | | Independent Adjudication Committee | |
| 16.2.8 | | Listing of Individual Laboratory | |
| | | Measurements by Subject | |
| 16.2.8.1 | | Clinical Laboratory Data | |
| | 16.2.8.1.1 | Laboratory Data - Hematology | Safety Population |
| | 16.2.8.1.2 | Laboratory Data - Clinical Chemistry | Safety Population |
| | 16.2.8.1.3 | Laboratory Data - Urinalysis | Safety Population |
| | 16.2.8.1.4 | Childbearing Potential and Premenses | Safety Population |
| | | Status | |
| | 16.2.8.1.5 | Pregnancy Test Results | Safety Population |
| | 16.2.8.1.6 | Tuberculosis Test Results | Safety Population |
| | 16.2.8.1.7 | Virology | Safety Population |
| 16.2.8.2 | | Other Safety Data | |
| | 16.2.8.2.1 | Vital Signs, Height and Weight | Safety Population |
| | 16.2.8.2.2 | Electrocardiogram (ECG) | Safety Population |

| | Listing | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| | 16.2.8.2.3 | Physical Examination | Safety Population |
| | 16.2.8.2.4 | Respiratory Assessment – Medical Interview | Safety Population |
| | 16.2.8.2.5 | Respiratory Assessment – Peak Expiratory Flow (PEF) | Safety Population |
| | 16.2.8.2.6 | Known Asthma, Wheeze, Dyspnea and Cough Triggers | Safety Population |
| | 16.2.8.2.7 | Asthma Control Test (ACT) | Safety Population |
| | 16.2.8.2.8 | Subjects with a drop by >= 15% from Baseline for either PEF or ACT | Safety Population |

#### 20. Appendices

#### 20.1. Example SAS Code

1. The Example SAS code for Time to Event and Hazard Ratio

```
proc lifetest data=analysis_data;
time aval*cnsr(1);
strata trtp;
run;
proc phreg data=analysis_data;
class trtp stratum;
model aval*cnsr(1)=trtp stratum;
run;
```

2. The example SAS code for CMH model is listed as below:

```
proc freq data=analysis_data;
tables stratum*trt*resp/ cmh alpha=0.1;
run;
```

3. The example SAS code for MMRM model is listed as below:

```
proc mixed data = analysis_data;

class stratum trtp avisit subjid;

model chg = base stratum trtp avisit trtp*avisit/ ddfm=kr;

repeated avisit / subject=subjid(trtp) type=un;

Ismeans trtp/ cl diff;

Ismeans trtp*avisit/ slice=avisit cl diff;

run;
```

4. The example SAS code for ANCOVA model is listed as below:

```
proc mixed data = analysis_data;

class stratum trtp;

model chg = base stratum trtp;
```

This document is confidential.

SAP Version: 2.0 19-Jan-2024

Controlled Document ID: 3903A.02, Effective Date 31-Aug-2020

Filing requirements: TMF

Statistical Analysis Plan for Interventional Studies

Ismeans trtp/ cl diff;

run;

### 20.2. Potentially Clinically Significant Ranges

Potentially clinically significant ranges for Hematology parameters are defined in Table 20-1.

Table 20-1 Potentially Clinically Significant Ranges for Hematology Parameters

| Test Parameter | Test<br>Parameter<br>Code | Normal Range Lower<br>Limit (LLN) | Normal Range Upper<br>Limit (ULN) | Potentially Clinically Significant Ranges |
|---|---|---|---|---|
| Basophils (x10^9/L) | BASO | 0.00 | 0.20 | > 0.2 at post-baseline, if baseline value ≤ 0.2 |
| Eosinophils (x10^9/L) | EOS | 0.00 | 0.57 | > 0.7 at post-baseline, if baseline value ≤ 0.7 |
| Hematocrit (L/L) | нст | 0.39 (12-<59 years old,<br>Male) | 0.54 (12-<59 years old, Male) | < 0.30 at post-baseline, if baseline value ≥ 0.30 |
| | | 0.37 (≥ 59 years old,<br>Male) | 0.51 (≥ 59 years old,<br>Male) | > 0.6 at post-baseline, if baseline value ≤ 0.6 |
| | | 0.34 (Female) | 158.00 (Female) | |
| Hemoglobin (g/L) | HGB | 127 (12-<59 years old,<br>Male) | 181 (12-<59 years old,<br>Male) | Male < 100 at post-baseline, if baseline value ≥ 100 |
| | | 116 (12-<59 years old,<br>Female) | 164 (12-<59 years old,<br>Female) | Male ≥ 200 at post-baseline, if baseline value < 200 |
| | | 125 (≥ 59 years old,<br>Male) | 170 (≥ 59 years old,<br>Male) | Female <90 g/L at post-baseline and ≥ 90 g/L at baseline |
| | | 115 (≥ 59 years old,<br>Female) | 158 (≥ 59 years old,<br>Female) | Female ≥180 g/L at post-baseline and < 180 g/L at baseline |
| Leukocytes (x10^9/L) | WBC | 3.80 | 10.70 | < 3.0 at post-baseline, if baseline value ≥ 3.0 |
| | | | | > 15.0 at post-baseline, if baseline value ≤ 15.0 |
| Lymphocytes (x10^9/L) | LYM | 0.91 (18 – <59 years old) | 4.28 (18 – <59 years old) | < 0.8 at post-baseline, if baseline value ≥ 0.8 |
| | | 0.80 (≥ 59 years old) | 3 (≥ 59 years old) | > 4.28 at post-baseline, if baseline value ≤ 4.28 (age 18 - < 59); > 3.00 at post-baseline, if baseline value ≤ 3.00 (age ≥ 59) |
| Monocytes (x10^9/L) | MONO | 0.12 | 0.92 | > 0.92 at post-baseline, if baseline value ≤ 0.92 |

| Neutrophils,<br>Segmented (GI/L) | NEUTSG | 1.96 | 7.23 | < 1.5 at post-baseline, if baseline value is ≥ 1.5 |
|---|---|---|---|---|
| | | | | > 9 at post-baseline, if baseline value is ≤ 9 |
| Platelets (x10^9/L) | PLAT | 140 (18 - <60 years old) | 400 (18 - <60 years old) | < 100 at post-baseline, if baseline value ≥ 100 |
| | | 130 (≥ 60 years old) | 394 (≥ 60 years old) | > 700 at post-baseline, if baseline value ≤ 700 |

Potentially clinically significant ranges for Blood Chemistry parameters are defined in Table 20-2 Potentially Clinically Significant Ranges for Blood Chemistry Parameters.

Table 20-2 Potentially Clinically Significant Ranges for Blood Chemistry Parameters

| Test Parameter | Test<br>Parameter<br>Code | Normal Range Lower<br>Limit (LLN) | Normal Range Upper<br>Limit (ULN) | Potentially Clinically Significant Ranges |
|---|---|---|---|---|
| Aspartate<br>Aminotransferase (U/L) | AST | 8.00 | 40.00 | > 3 x ULN at post-baseline, if baseline value ≤ 3 x ULN |
| Alkaline Phosphatase (U/L) | ALP | 55 (< 19 years old,<br>Male) | 149 (< 19 years old,<br>Male) | > 2.5 x ULN at post-baseline, if baseline value ≤ 2.5 x ULN |
| | | 45 (< 19 years old,<br>Female) | 87 (< 19 years old,<br>Female) | |
| | | 40 (≥ 19 years old,<br>Male) | 129(≥ 19 years old,<br>Male) | |
| | | 35 (≥ 19 years old,<br>Female) | 104 (≥ 19 years old,<br>Female) | |
| Alanine<br>Aminotransferase (U/L) | ALT | 5 (Male) | 48 (Male) | > 3 x ULN at post-baseline, if baseline value ≤ 3 x ULN |
| | | 4 (Female) | 43 (Female) | |
| Bilirubin (umol/L) | BILI | 3.00 | 21.00 | > 1.5 x ULN at post-baseline, if baseline value ≤ 1.5 * ULN |
| Calcium (mmol/L) | CA | 2.07 | 2.64 | < 2 at post-baseline, if baseline value ≥ 2 |
| | | | | > 2.9 at post-baseline, if baseline value ≤ 2.9 |
| Chloride (mmol/L) | CL | 94.00 | 112.00 | < 94 at post-baseline, if baseline value ≥ 94 |
| | | | | > 115 at post-baseline, if baseline value ≤ 115 |
| Cholesterol (mmol/L) | CHOL | 2.95 (< 20 years old,<br>Male) | 5.12 (< 20 years old,<br>Male) | > 7.75 at post-baseline, if baseline value ≤ 7.75 (Female ≤ 60 years old, Male ≤ 70 years old); > 8.28 at post-baseline, if baseline value ≤ 8.28 (Female < 60 - 70 years old); > 7.76 at post-baseline, if baseline value ≤ 7.76 (Male > 70 years old); > 9.10 at post-baseline, if baseline value ≤ 9.10 (Female > 70 years old) |
| | | 3.23 (< 20 years old, Female) | 5.48 (< 20 years old,<br>Female) | |

| Test Parameter | Test<br>Parameter<br>Code | Normal Range Lower<br>Limit (LLN) | Normal Range Upper<br>Limit (ULN) | Potentially Clinically Significant Ranges |
|---|---|---|---|---|
| | | 3.31 (20 - < 30 years | 6.10 (20 - < 30 years | |
| | | old, Male) | old, Male) | |
| | | 3.31 (20 - < 30 years | 5.64 (20 - < 30 years old, Female) | |
| | | old, Female)<br>3.88 (30 - < 40 years | 6.83 (30 - < 40 years | |
| | | old, Male) | old, Male) | |
| | | 3.65 (30 - < 40 years | 6.21 (30 - < 40 years | |
| | | old, Female) | old, Female) | |
| | | 4.19 (40 - < 50 years | 7.24 (40 - < 50 years | |
| | | old, Male) | old, Male) | |
| | | 4.01 (40 - < 50 years | 6.85 (40 - < 50 years | |
| | | old, Female) | old, Female) | |
| | | 4.40 (50 - < 60 years | 7.53 (50 - < 60 years | |
| | | old, Male) | old, Male) | |
| | | 4.42 (50 - < 60 years | 7.53 (50 - < 60 years | |
| | | old, Female) | old, Female) | |
| | | 4.53 (60 - < 70 years | 7.71 (60 - < 70 years | |
| | | old, Male) | old, Male) | |
| | | 4.86 (60 - < 70 years | 8.28 (60 - < 70 years | |
| | | old, Female) | old, Female) | |
| | | 4.58 (≥ 70 years old, Male) | 7.76 (≥ 70 years old,<br>Male) | |
| | | 5.35 (≥ 70 years old, | 9.10 (≥ 70 years old, | |
| | | Female) | Female) | |
| Creatinine (umol/L) | CREAT | 40 (18 - < 50 years | 110 (18 - < 50 years | > 1.5 x ULN at post-baseline, if baseline value ≤ 1.5 |
| | | old, Male) | old, Male) | x ULN |
| | | 31 (18 - < 50 years | 101 (18 - < 50 years | |
| | | old, Female) | old, Female) | |
| | | 40 (50 - < 70 years | 119 (50 - < 70 years | |
| | | old, Male) | old, Male) | |
| | | 31 (50 - < 70 years | 101 (50 - < 70 years | |
| | | old, Female) | old, Female) | |
| | | 40 (70 - < 80 years | 137 (70 - < 80 years | |
| | | old, Male) | old, Male) | |

| Test Parameter | Test<br>Parameter<br>Code | Normal Range Lower<br>Limit (LLN) | Normal Range Upper<br>Limit (ULN) | Potentially Clinically Significant Ranges |
|---|---|---|---|---|
| | | 31 (70 - < 80 years | 110 (70 - < 80 years | |
| | | old, Female) | old, Female) | |
| | | 40 (≥ 80 years old, | 145 (≥ 80 years old, | |
| | | Male) | Male) | |
| | | 31 (≥ 80 years old,<br>Female) | 128 (≥ 80 years old,<br>Female) | |
| Creatine Kinase (U/L) | CK | 39 (Male) | 308 (Male) | > 2.5 x ULN at post-baseline, if baseline value ≤ 2.5 x ULN |
| | | 26 (Female) | 192 (Female) | |
| Direct Bilirubin (umol/L) | BILDIR | <2.00 | 7.00 | > 1.5 x ULN at post-baseline, if baseline value ≤ 1.5 x ULN |
| Gamma Glutamyl<br>Transferase (U/L) | GGT | 10 (< 59 years old,<br>Male) | 61 (< 59 years old,<br>Male) | > 2.5 x ULN at post-baseline, if baseline value ≤ 2.5 x ULN |
| | | 4 (< 59 years old,<br>Female) | 49 (< 59 years old,<br>Female) | |
| | | 10 (≥ 59 years old,<br>Male) | 50 (≥ 59 years old,<br>Male) | |
| | | 5 (≥ 59 years old,<br>Female) | 50 (≥ 59 years old,<br>Female) | |
| Glucose (mmol/L) | GLUC | 3.90 | 5.60 | < 3 at post-baseline, if baseline value ≥ 3 |
| • | | | | > 13.9 at post-baseline, if baseline value ≤ 13.9 |
| Potassium (mmol/L) | K | 3.5 | 5.2 | < 3.5 at post-baseline, if baseline value ≥ 3.5 |
| , | | | | > 5.5 at post-baseline, if baseline value ≤ 5.5 |
| Sodium (mmol/L) | SODIUM | 132 (18 – < 59 years old) | 147 (18 – < 59 years old) | < 129 at post-baseline, if baseline value ≥ 129 |
| | | 135 (≥ 59 years old) | 145 (≥ 59 years old) | > 150 at post-baseline, if baseline value ≤ 150 |
| Triglycerides (mmol/L) | TRIG | 0.42 (< 20 years old,<br>Male) | 1.67 (< 20 years old,<br>Male) | > 3.69 at post-baseline, if baseline value ≤ 3.69 |
| | | 0.44 (< 20 years old,<br>Female) | 1.40 (< 20 years old,<br>Female) | |
| | | 0.50 (20 – < 30 years old, Male) | 2.81 (20 – < 30 years old, Male) | |
| | | 0.41 (20 – < 30 years old, Female) | 1.63 (20 – < 30 years old, Female) | |

| Test Parameter | Test<br>Parameter<br>Code | Normal Range Lower<br>Limit (LLN) | Normal Range Upper<br>Limit (ULN) | Potentially Clinically Significant Ranges |
|---|---|---|---|---|
| | | 0.56 (30 – < 40 years old, Male) | 3.62 (30 – < 40 years old, Male) | |
| | | 0.44 (30 <b>–</b> < 40 years | 1.99 (30 – < 40 years | |
| | | old, Female) | old, Female) | |
| | | 0.62 (40 <b>–</b> < 50 years old, Male) | 3.69 (40 <b>–</b> < 50 years old, Male) | |
| | | 0.51 (40 – < 50 years | 2.42 (40 – < 50 years | |
| | | old, Female)<br>0.65 (50 – < 60 years<br>old, Male) | old, Female)<br>3.61 (50 – < 60 years<br>old, Male) | |
| | | 0.59 (50 – < 60 years old, Female) | 2.96 (50 – < 60 years old, Female) | |
| | | 0.65 (≥ 60 years old,<br>Male) | 2.94 (≥ 60 years old,<br>Male) | |
| | | 0.63 (≥ 60 years old,<br>Female) | 2.71 (≥ 60 years old,<br>Female) | |
| Urate (mmol/L) | URATE | 125 (< 50 years old,<br>Male) | 488 (< 50 years old,<br>Male) | > 494 at post-baseline, if baseline value ≤ 494 (Male);<br>> 446 at post-baseline, if baseline value ≤ 446 (Female) |
| | | 125 (< 50 years old,<br>Female) | 428 (< 50 years old,<br>Female) | |
| | | 149 (50 - < 70 years old, Male) | 494 (50 - < 70 years old, Male) | |
| | | 149 (50 - <70 years old, Female) | 446 (50 - < 70 years old, Female) | |
| | | 149 (≥ 70 years old,<br>Male) | 494 (≥ 70 years old,<br>Male) | |
| | | 149 (≥ 70 years old,<br>Female) | 446 (≥ 70 years old,<br>Female) | |
| Urea Nitrogen (mmol/L) | UREAN | 1.40 (< 70 years old) | 8.60 (< 70 years old) | > 8.6 at post-baseline, if baseline value ≤ 8.6 (<70 years old); > 10.4 at post-baseline, if baseline value ≤ 10.4 (70 - <80 years old); > 12.1 at post-baseline, if baseline value ≤ 12.1 (≥ 80 years old) |

Statistical Analysis Plan for Interventional Studies

| Test Parameter | Test<br>Parameter<br>Code | Normal Range Lower<br>Limit (LLN) | Normal Range Upper<br>Limit (ULN) | Potentially Clinically Significant Ranges |
|---|---|---|---|---|
| | | 1.40 (70 - < 80 years | 10.40 (70 - < 80 years | |
| | | old) | old) | |
| | | 1.40 (≥ 80 years old) | 12.10 (≥ 80 years old) | |

Potentially clinically significant ranges for vital signs parameters are defined in Table 20-3.

Table 20-3 Potentially Clinically Significant Ranges for Vital Signs Parameters

| Test Parameter | Test Parameter Code | Potentially Clinically Significant Ranges |
|---|---|---|
| Pulse rate (beats/min) | PULSE | ≥120 bpm and increase from baseline ≥20 bpm |
| | | ≤50 bpm and decrease from baseline ≥20 bpm |
| Diastolic blood pressure (mmHg) | DIABP | ≥110 mmHg and increase from baseline ≥10 mmHg |
| | | ≤45 mmHg and decrease from baseline ≥10 mmHg |
| Systolic blood pressure (mmHg) | SYSBP | ≥160 mmHg and increase from baseline ≥20 mmHg |
| | | ≤95 mmHg and decrease from baseline ≥20 mmHg |
| Weight | WEIGHT | ≥5% increase from baseline |
| | | ≥5% decrease from baseline |



